CLINICAL TRIAL: NCT03191786
Title: A Phase III, Open-Label, Multicenter, Randomized Study to Investigate the Efficacy and Safety of Atezolizumab Compared With Chemotherapy in Patients With Treatment Naïve Advanced or Recurrent (Stage IIIb Not Amenable for Multimodality Treatment) or Metastatic (Stage IV) Non-Small Cell Lung Cancer Who Are Deemed Unsuitable for Platinum-Containing Therapy
Brief Title: A Study of Atezolizumab Compared With a Single-Agent Chemotherapy in Treatment Naïve Participants With Locally Advanced or Recurrent or Metastatic Non-Small Cell Lung Cancer Who Are Deemed Unsuitable For Platinum-Doublet Chemotherapy
Acronym: IPSOS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MO29872; 2015-004105-16 (EudraCT Number)
Record Dates: First submitted 2017-06-15; First posted 2017-06-19 (Actual); Results first posted 2023-05-17 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2024-09

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — atezolizumab; Vinorelbine; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Atezolizumab (Experimental): Participants will receive atezolizumab 1200 milligrams (mg) intravenous (IV) infusion on Day 1 of each 21-day cycle until loss of clinical benefit, unacceptable toxicity, participant or physician decision to discontinue, or death.
  Interventions: Drug: Atezolizumab (MPDL3280A), an engineered anti-PD-L1 antibody
- Single Agent Chemotherapy (Vinorelbine or Gemcitabine) (Active Comparator): Participants will receive single agent chemotherapy; either vinorelbine oral or IV, or gemcitabine IV, according to the label based on investigator's choice.
  Interventions: Drug: Vinorelbine; Drug: Gemcitabine

INTERVENTIONS:
Drug: Atezolizumab (MPDL3280A), an engineered anti-PD-L1 antibody — Atezolizumab will be administered via IV infusion once every three weeks (QW3).
  Other Names: MPDL3280A
  Arms: Atezolizumab
Drug: Vinorelbine — Vinorelbine will be administered per relevant local guidelines and Summary of Product Characteristics (SmPC) management.
  Other Names: Navelbine®
  Arms: Single Agent Chemotherapy (Vinorelbine or Gemcitabine)
Drug: Gemcitabine — Gemcitabine will be administered per relevant local guidelines and SmPC management.
  Other Names: Gemzar®
  Arms: Single Agent Chemotherapy (Vinorelbine or Gemcitabine)

SUMMARY:
This Phase III, global, multicenter, open-label, randomized, controlled study will evaluate the efficacy and safety of atezolizumab (an anti-programmed death-ligand 1 [anti-PD-L1] antibody) compared with a single agent chemotherapy regimen by investigator choice (vinorelbine or gemcitabine) in treatment-naïve participants with locally advanced or metastatic non-small cell lung cancer (NSCLC) who are deemed unsuitable for any platinum-doublet chemotherapy due to poor performance status (Eastern Cooperative Oncology Group [ECOG] performance status of 2-3).

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed diagnosis of advanced or recurrent (Stage IIIB not amenable for multimodality treatment) or metastatic (Stage IV) NSCLC as per the American Joint Committee on Cancer (AJCC) 7th edition
* No sensitizing epidermal growth factor receptor (EGFR) mutation (L858R or exon 19 deletions) or anaplastic lymphoma kinase (ALK) fusion oncogene detected
* No prior systemic treatment for advanced or recurrent (Stage IIIB not amenable for multimodality treatment) or metastatic (Stage IV) NSCLC as per the AJCC 7th edition
* Life expectancy greater than or equal to (>/=) 8 weeks
* Deemed unsuitable by the investigator for any platinum-doublet chemotherapy due to poor performance status (ECOG performance status of 2-3). However, participants >= 70 years of age who have an ECOG PS of 0 or 1 may be included due to: a) substantial comorbidities; b) contraindication(s) for any platinum-doublet chemotherapy
* Representative formalin-fixed paraffin-embedded (FPPE) tumor tissue block obtained during course of disease (archival tissue) or at screening
* Participants with treated, asymptomatic central nervous system (CNS) metastases are eligible, provided they meet all of the following criteria: Measurable disease outside CNS; Only supratentorial and cerebellar metastases allowed; No ongoing requirement for corticosteroids as therapy for CNS disease; No stereotactic radiation within 7 days or whole-brain radiation within 14 days prior to randomization; No evidence of interim progression between the completion of CNS-directed therapy and the screening radiographic study
* Adequate hematologic and end organ function
* Female participants of childbearing potential randomized to the atezolizumab treatment arm agree to use protocol defined methods of contraception

Exclusion Criteria:

Cancer-Specific Exclusion Criteria:

* Participants younger than 70 years who have an ECOG performance status of 0 or 1
* Active or untreated CNS metastases as determined by computed tomography (CT) or magnetic resonance imaging (MRI) evaluation of the brain during screening and prior radiographic assessments
* Uncontrolled tumor-related pain
* Uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures (once monthly or more frequently)
* Uncontrolled or symptomatic hyerpcalcemia (ionized calcium > 1.5 mmol/L or calcium >12 mg/dL or corrected serum calcium >ULN)
* History of other malignancy within 5 years prior to screening, with the exception of those with a negligible risk of metastasis or death treated with expected curative outcome
* National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 4.0 (v4.0) Grade 3 or higher toxicities due to any prior therapy (example [e.g.], radiotherapy) (excluding alopecia), which have not shown improvement and are strictly considered to interfere with current study medication
* Participants who have received prior neo-adjuvant, adjuvant chemotherapy, radiotherapy, or chemoradiotherapy with curative intent for non-metastatic disease must have experienced a treatment-free interval of at least 6 months from randomization since the last chemotherapy, radiotherapy, or chemoradiotherapy

General Medical Exclusion Criteria:

* History of autoimmune disease except autoimmune-related hypothyroidism and controlled Type I diabetes mellitus
* History of idiopathic pulmonary fibrosis (IPF), organizing pneumonia (e.g., bronchiolitis obliterans), drug-induced pneumonitis, idiopathic pneumonitis, or evidence of active pneumonitis
* Known positivity for human immunodeficiency virus (HIV)
* Known active hepatitis B or hepatitis C
* Active tuberculosis
* Severe infections within 4 weeks prior to randomization
* Significant cardiovascular disease, such as New York Heart Association (NYHA) cardiac disease (Class II or greater), myocardial infarction within 3 months prior to randomization, unstable arrhythmias, or unstable angina
* Major surgical procedure other than for diagnosis within 4 weeks prior to randomization or anticipation of need for a major surgical procedure during the course of the study
* Prior allogeneic bone marrow transplantation or solid organ transplant
* Participants with an illness or condition that may interfere with capacity or compliance with the study protocol, as per investigator's judgment
* Treatment with any other investigational agent or participation in another clinical study with therapeutic intent within 28 days prior to randomization

Exclusion Criteria Related to Atezolizumab:

* History of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric or humanized antibodies or fusion proteins
* Known hypersensitivity to biopharmaceuticals produced in Chinese hamster ovary cells or any component of the atezolizumab formulation
* Oral or IV antibiotic treatment
* Administration of a live, attenuated vaccine within 4 weeks before randomization or anticipation that such a live attenuated vaccine will be required during the study
* Prior treatment with cluster of differentiation 137 (CD137) agonists or immune checkpoint blockade therapies, anti-programmed death-1 (anti-PD-1), and anti-PD-L1 therapeutic antibodies
* Treatment with systemic immunostimulatory agents within 4 weeks or 5 half-lives of the drug, whichever is shorter, prior to randomization
* Treatment with systemic corticosteroids or other immunosuppressive medications
* Participants not willing to stop treatment with traditional herbal medicines

Exclusion Criteria Related to Chemotherapy:

* Known sensitivity and contraindications to the 2 comparative chemotherapy agents (that is [i.e.] vinorelbine, oral or intravenous, and gemcitabine, intravenous)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 453 (Actual)
Dates: Start 2017-09-11 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2023-10-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (91):
- Argentina (3):
  - Fundación CENIT para la Investigación en Neurociencias, Buenos Aires
  - Hospital Privado de Comunidad, Mar del Plata
  - Clinica Viedma S.A., Viedma
- Belgium (3):
  - UZ Brussel, Brussels
  - Grand Hôpital de Charleroi Notre Dame, Charleroi
  - UZ Leuven Gasthuisberg, Leuven
- Brazil (3):
  - Hospital Nossa Senhora da Conceicao, Porto Alegre, Rio Grande do Sul
  - Hospital Sao Lucas - PUCRS, Porto Alegre, Rio Grande do Sul
  - Instituto do Cancer do Estado de Sao Paulo - ICESP, São Paulo, São Paulo
- Bulgaria (2):
  - Umhat Dr Georgi Stranski; Clinic of Chemotherapy, Pleven
  - Complex Oncology Center (COC)-Plovidiv, Plovdiv
- Canada (5):
  - BCCA-Vancouver Cancer Centre, Vancouver, British Columbia
  - Regional health authority A vitalite health network, Moncton, New Brunswick
  - Ottawa Hospital Research Institute, Ottawa, Ontario
  - Princess Margaret Cancer Center, Toronto, Ontario
  - Jewish General Hospital, Montreal, Quebec
- China (7):
  - Beijing Cancer Hospital, Beijing
  - Hu Nan Provincial Cancer Hospital, Changsha
  - The Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou
  - Anhui Provincial Hospital, Hefei
  - Shanghai Chest Hospital, Shanghai
  - Tianjin Cancer Hospital, Tianjin
  - Union Hospital of Tongji Medical College, Dept. of Cancer Center; Cancer Center, Wuhan
- Colombia (4):
  - Fundacion Cardioinfantil, Bogotá
  - Fundación Centro de Investigación Clínica CIC, Medellín
  - Oncomedica S.A., Montería
  - Oncólogos de Occidente, Pereira
- Fakultni nemocnice Olomouc; Pneumologicka klinika, Olomouc, Czechia
- Odense Universitetshospital, Onkologisk Afdeling R, Odense C, Denmark
- Germany (8):
  - Evang. Lungenklinik Berlin Klinik für Pneumologie, Berlin
  - Asklepios Klinik Gauting; Onkologisches Studienzentrum, Gauting
  - LungenClinic Großhansdorf GmbH; Klinische Forschung, Großhansdorf
  - Krankenhaus Martha-Maria Halle-Doelau gGmbH; Klinik fuer Innere Medizin II, Halle
  - Fachklinik für Lungenerkrankungen, Immenhausen
  - Klinikum der Philipps-Universität Marburg, Marburg
  - Universitätsklinikum Regensburg; Klinik und Poliklinik für Innere Medizin II, Pneumologie, Regensburg
  - Universitätsklinikum Tübingen; Innere Medizin VIII, Medizinische Onkologie und Pneumologie, Tübingen
- India (13):
  - HealthCare Global Cancer Centre; Medical Oncology, Ahmedabad, Gujarat
  - Kailash Cancer Hospital and Research Center, Vadodara, Gujarat
  - P.D. Hinduja Nat. Hospital & Med. Research Centre, Mahim(West), Maharashtra
  - Tata Memorial Hospital; Dept of Medical Oncology, Mumbai, Maharashtra
  - Kokilaben Dhirubhai Ambani Hospital & Medical Research Institute; Department of Rheumatologz, Mumbai, Maharashtra
  - HCG Manavata Cancer Centre, Nashik, Maharashtra
  - Grant Medical Foundation, Ruby Hall Clinic, Pune, Maharashtra
  - Deenanath Mangeshkar Hospital & Research Centre, Pune, Maharashtra
  - Max Super Speciality Hospital, New Delhi, National Capital Territory of Delhi
  - Indraprastha Apollo Hospitals, New Delhi, National Capital Territory of Delhi
  - Rajiv Gandhi Cancer Inst.&Research Center; Medical Oncology, New Delhi, National Capital Territory of Delhi
  - Indo-American Cancer Hospital & Research Center, Hyderabad, Telangana
  - Tata Medical Center; Department of Medical Oncology, Kolkata, West Bengal
- Ireland (2):
  - Mater Misericordiae University Hospital - Institute for Cancer Research, Dublin
  - University Hospital Limerick - Clinical Trials Department, Limerick
- Italy (3):
  - Ospedale Provinciale Santa Maria Delle Croci; Oncologia Medica, Ravenna, Emilia-Romagna
  - Azienda Ospedaliera San Camillo Forlanini; U.O.C. Pneumologia Ad Indirizzo Oncologico 1, Rome, Lazio
  - Azienda Ospedaliera San Gerardo di Monza, Monza MI, Lombardy
- Kazakhstan (2):
  - Kazakh Scientific Research Institution Of Oncology and Radiology, Almaty
  - Almaty Oncology Center, Almaty
- Centre Hospitalier de Luxembourg, Luxembourg, Luxembourg
- Mexico (3):
  - Health Pharma Professional Research, Mexico City, Mexico CITY (federal District)
  - Oncologico Potosino, San Luis Potosí City, San Luis Potosí
  - Centro Estatal de Cancerologia de Chihuahua; ONCOLOGY, Chihuahua City
- Poland (2):
  - Mazowieckie Centrum Leczenia Chorob Pluc I Gruzlicy; Oddzial Iii, Otwock
  - Narod.Inst.Onkol. im. M.Sklodowskiej - Curie-Panst.Inst.Bad; Klinika Nowot.Pluca i Klatki Piers, Warsaw
- Portugal (2):
  - CHUC - Unidade de Pneumologia Oncológica; Hospital de Dia de Oncologia Edificio Sao Jeronimo, Coimbra
  - IPO do Porto; Servico de Oncologia Medica, Porto
- Romania (3):
  - Institutul Oncologic Prof. Dr. Ion Chiricuta Cluj Napoca; Oncologie Medicala, Cluj-Napoca
  - Centrul de Radioterapie AMETHYST, Floreşti
  - Oncocenter Timisoara, Timi?oara
- Slovakia (2):
  - Specializovana nemocnica sv. Svorada Zobor, n.o.; Oddelenie klinickej onkologie, Nitra
  - Fakultna nemocnica Trnava, Trnava
- Spain (9):
  - Complejo Hospitalario Universitario de Santiago (CHUS) ; Servicio de Oncologia, Santiago de Compostela, LA Coruña
  - Hospital de Cruces; Servicio de Oncologia, Bilbao, Vizcaya
  - Institut Catala d Oncologia Hospital Duran i Reynals, Barcelona
  - Hospital Universitario de la Princesa; Servicio de Oncologia, Madrid
  - Hospital Universitario Clínico San Carlos; Servicio de Oncologia, Madrid
  - Hospital Clinico Universitario Virgen de la Victoria; Servicio de Oncologia, Málaga
  - Hospital General Universitario J.M Morales Meseguer; Servicio de Oncologia, Murcia
  - Hospital Universitario Virgen Macarena; Servicio de Oncologia, Seville
  - Hospital Arnau de Vilanova (Valencia) Servicio de Oncologia, Valencia
- Switzerland (3):
  - Ospedale Regionale di Bellinzona Medizin Onkologie, Bellinzona
  - Spital STS AG - Spital Thun Medizin Onkologie; MEDIZINISCHE KLINIK, Thun
  - Kantonsspital Winterthur; Medizinische Onkologie, Winterthur
- United Kingdom (7):
  - Clatterbridge Cancer Centre, Bebington
  - Birmingham Heartlands Hospital, Birmingham
  - Royal Cornwall Hospital; Dept of Clinical Oncology, Cornwall
  - New Victoria Hospital, Glasgow
  - University College London Hospitals NHS Foundation Trust - University College Hospital, London
  - Christie Hospital Nhs Trust; Medical Oncology, Manchester
  - YORK DISTRICT HOSPITAL; Haematology/Oncology Department, York
- Vietnam (2):
  - Bach Mai Hospital, Hanoi
  - Cho Ray Hospital, Hochiminh City

REFERENCES:
- [Derived] Han B, Peters S, Le AT, Huang D, Wu G, Cao L, Pham CP, Zhao J, Wang K, Yang N, Zhong H, Hu Y, Morris S, Lam V, Graupner V, Gitlitz B, Hoglander E, Schulz C, Lee SM. First-line atezolizumab monotherapy vs. single-agent chemotherapy in patients with advanced or metastatic non-small cell lung cancer who are ineligible for platinum-based therapy: Analysis of the IPSOS Asian subpopulation. Chin Med J (Engl). 2025 Dec 17. doi: 10.1097/CM9.0000000000003796. Online ahead of print. PMID 41424028
- [Derived] Li B, Rong D, Lin H. Atezolizumab monotherapy as first-line treatment for non-small cell lung cancer ineligible for treatment with a platinum-containing regimen (IPSOS): a cost-effectiveness analysis in the USA. BMJ Open. 2024 Nov 12;14(11):e083716. doi: 10.1136/bmjopen-2023-083716. PMID 39532375
- [Derived] Lee SM, Schulz C, Prabhash K, Kowalski D, Szczesna A, Han B, Rittmeyer A, Talbot T, Vicente D, Califano R, Cortinovis D, Le AT, Huang D, Liu G, Cappuzzo F, Reyes Contreras J, Reck M, Palmero R, Mak MP, Hu Y, Morris S, Hoglander E, Connors M, Biggane AM, Vollan HK, Peters S. First-line atezolizumab monotherapy versus single-agent chemotherapy in patients with non-small-cell lung cancer ineligible for treatment with a platinum-containing regimen (IPSOS): a phase 3, global, multicentre, open-label, randomised controlled study. Lancet. 2023 Aug 5;402(10400):451-463. doi: 10.1016/S0140-6736(23)00774-2. Epub 2023 Jul 6. PMID 37423228
- [Derived] Gijtenbeek RG, de Jong K, Venmans BJ, van Vollenhoven FH, Ten Brinke A, Van der Wekken AJ, van Geffen WH. Best first-line therapy for people with advanced non-small cell lung cancer, performance status 2 without a targetable mutation or with an unknown mutation status. Cochrane Database Syst Rev. 2023 Jul 7;7(7):CD013382. doi: 10.1002/14651858.CD013382.pub2. PMID 37419867

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants diagnosed with advanced or recurrent (stage IIIb) or metastatic (stage IV) non-small cell lung cancer (NSCLC) took part in the study across 85 investigative sites in 23 countries from 11 Sep 2017 to 25 Oct 2023.
Pre-assignment Details: A total of 453 participants were randomized in 2:1 ratio to atezolizumab arm and single agent chemotherapy arm(vinorelbine or gemcitabine) in this study. 447 participants received at least one dose of study treatment.
Groups:
- Atezolizumab: Participants received atezolizumab 1200 milligrams (mg), as intravenous (IV) infusion on Day 1 of each 21-day cycle until loss of clinical benefit, unacceptable toxicity, participant or physician decision to discontinue, or death.
- Single Agent Chemotherapy (Vinorelbine or Gemcitabine): Participants received single agent chemotherapy; either vinorelbine oral or IV, or gemcitabine IV, according to the label based on investigator's choice until disease progression unacceptable toxicity, participant or physician decision to discontinue, or death.
Period: Overall Study
Arm/Group | Atezolizumab | Single Agent Chemotherapy (Vinorelbine or Gemcitabine)
Started | 302 | 151
Safety Evaluable Population (Safety-evaluable population included all randomized participants who received any amount of study treatment.) | 300 | 147
Completed | 0 | 0
Not Completed | 302 | 151
Not completed — Death | 236 | 127
Not completed — Lost to Follow-up | 9 | 3
Not completed — Physician Decision | 1 | 0
Not completed — Moved to Post Trial Access Program | 30 | 5
Not completed — Withdrawal by Subject | 26 | 16

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population included all randomized participants irrespective of whether the assigned treatment was actually received.
Groups:
- Atezolizumab: Participants received atezolizumab 1200 mg, as IV infusion on Day 1 of each 21-day cycle until loss of clinical benefit, unacceptable toxicity, participant or physician decision to discontinue, or death.
- Total: Total of all reporting groups
Arm/Group | Atezolizumab | Single Agent Chemotherapy (Vinorelbine or Gemcitabine) | Total
Number analyzed (Participants) | 302 | 151 | 453
Age, Continuous [Mean (Standard Deviation); unit: Years] | 73.6 (9.1) | 73.8 (8.5) | 73.7 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 82 | 43 | 125
  Male | 220 | 108 | 328
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 47 | 22 | 69
  Not Hispanic or Latino | 242 | 126 | 368
  Unknown or Not Reported | 13 | 3 | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 12 | 9 | 21
  Asian | 75 | 38 | 113
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 203 | 95 | 298
  More than one race | 6 | 6 | 12
  Unknown or Not Reported | 4 | 2 | 6

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS)
Description: OS was defined as the time between the date of randomization and the date of death due to any cause. Kaplan-Meier (KM) estimates were used to calculate median.
Time Frame: From randomization up to death from any cause (up to approximately 55 months)
Population: ITT population included all randomized participants irrespective of whether the assigned treatment was actually received.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Atezolizumab | Single Agent Chemotherapy (Vinorelbine or Gemcitabine)
Number analyzed (Participants) | 302 | 151
Months | 10.3 [9.4 to 11.9] | 9.2 [5.9 to 11.2]
Statistical Analysis 1: Comparison: Atezolizumab vs Single Agent Chemotherapy (Vinorelbine or Gemcitabine); Stratified analysis. Histologic subtype, PD-L1 IHC status and brain metastases (Yes/No) were added as stratification factors; Test type: Superiority; p = 0.025, Log Rank; Hazard Ratio (HR) = 0.78, 95% CI 2-sided [0.63 to 0.97]

2. Secondary Outcome: OS Rates at the 6, 12, 18, 24-Months Timepoints
Description: OS was defined as the time between the date of randomization and the date of death due to any cause. OS rate at 6, 12, 18 and 24 months were estimated for each treatment arm using Kaplan Meier methodology. Percentages were rounded off to the nearest decimal point.
Time Frame: 6, 12, 18 and 24 months
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Atezolizumab | Single Agent Chemotherapy (Vinorelbine or Gemcitabine)
Number analyzed (Participants) | 302 | 151
Percentage of participants
  6 Months | 64.0 [58.6 to 69.5] | 57.5 [49.4 to 65.7]
  12 Months | 43.7 [37.9 to 49.4] | 38.6 [30.5 to 46.7]
  18 Months | 31.4 [26.0 to 36.8] | 24.0 [16.8 to 31.2]
  24 Months | 24.3 [19.3 to 29.4] | 12.4 [6.7 to 18.0]
Statistical Analysis 1: Comparison: Atezolizumab vs Single Agent Chemotherapy (Vinorelbine or Gemcitabine); OS Rate at 6 Months; Test type: Superiority; Difference in OS Rates = 6.5, 95% CI 2-sided [-3.3 to 16.3]
Statistical Analysis 2: Comparison: Atezolizumab vs Single Agent Chemotherapy (Vinorelbine or Gemcitabine); OS Rate at 12 Months; Test type: Superiority; Difference in OS Rates = 5.1, 95% CI 2-sided [-4.9 to 15.0]
Statistical Analysis 3: Comparison: Atezolizumab vs Single Agent Chemotherapy (Vinorelbine or Gemcitabine); OS Rate at 18 Months; Test type: Superiority; Difference in OS Rates = 7.4, 95% CI 2-sided [-1.6 to 16.5]
Statistical Analysis 4: Comparison: Atezolizumab vs Single Agent Chemotherapy (Vinorelbine or Gemcitabine); OS Rate at 24 Months; Test type: Superiority; Difference in OS Rates = 11.9, 95% CI 2-sided [4.4 to 19.5]

3. Secondary Outcome: Percentage of Participants With Objective Response, as Determined by the Investigator Using Response Evaluation Criteria In Solid Tumors Version 1.1 (RECIST v1.1)
Description: Objective response rate (ORR)=best overall response (BOR) of either complete response (CR)/partial response (PR), as determined by investigator with use of RECIST v1.1. CR= disappearance of all target lesions or any pathological lymph nodes (whether target or non-target) having a reduction in short axis to <10 millimeters (mm). PR=at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum of diameters. A minimum interval of 6 weeks (42 days) was considered for stable disease (SD) to be assigned as BOR, i.e. in case the single response is SD, PR or CR, this single response must have been assessed no less than 6 weeks (at least 42 days) after start date of study treatment. SD=neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum of the diameters while in the study. Percentages were rounded off to the nearest decimal point.
Time Frame: From randomization to the first occurence of disease progression or death from any cause, whichever occurs first (up to approximately 55 months)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Atezolizumab | Single Agent Chemotherapy (Vinorelbine or Gemcitabine)
Number analyzed (Participants) | 302 | 151
Percentage of participants | 16.9 [12.8 to 21.6] | 7.9 [4.2 to 13.5]

4. Secondary Outcome: Progression-Free Survival (PFS), as Determined by the Investigator Using RECIST v1.1
Description: PFS was defined as the time from randomization to the first documented disease progression as determined by the investigator with the use of RECIST v1.1 or death from any cause, whichever occurs first. Progressive disease (PD) was defined as at least 20% increase in the sum of diameters of lesions, taking as reference the smallest sum during the study (nadir), including baseline. KM estimates were used to calculate median.
Time Frame: as for outcome 3
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Atezolizumab | Single Agent Chemotherapy (Vinorelbine or Gemcitabine)
Number analyzed (Participants) | 302 | 151
Months | 4.2 [3.7 to 5.5] | 4.0 [2.9 to 5.4]
Statistical Analysis 1: Comparison: Atezolizumab vs Single Agent Chemotherapy (Vinorelbine or Gemcitabine); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.182, Log Rank; Hazard Ratio (HR) = 0.87, 95% CI 2-sided [0.70 to 1.07]

5. Secondary Outcome: Duration of Response (DOR), as Determined by the Investigator Using RECIST v1.1
Description: DOR was defined as the time from the first tumor assessment that supports the participants' objective response (CR or PR, whichever is first reported) to documented disease progression as determined by the investigator according to RECIST v1.1 or death from any cause, whichever occurs first, among participants who have a best overall response as CR or PR. CR was defined as the disappearance of all target lesions or any pathological lymph nodes (whether target or non-target) having a reduction in short axis to <10 mm. PR was defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum of diameters. PD was defined as at least 20% increase in the sum of diameters of lesions, taking as reference the smallest sum during the study (nadir), including baseline. KM estimates were used to calculate median.
Time Frame: Time from the first occurrence of a documented objective response to the time of disease progression or death from any cause, whichever occurs first (up to approximately 55 months)
Population: ITT population included all randomized participants irrespective of whether the assigned treatment was actually received. Overall number analyzed is the number of participants with objective response (i.e. responders).
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Atezolizumab | Single Agent Chemotherapy (Vinorelbine or Gemcitabine)
Number analyzed (Participants) | 51 | 12
Months | 14.0 [8.1 to 20.3] | 7.8 [4.8 to 9.7]

6. Secondary Outcome: Percentage of Participants With At Least One Adverse Event (AE)
Description: An AE was any untoward medical occurrence in participant administered a pharmaceutical product & regardless of causal relationship with this treatment. An AE can therefore be any unfavorable & unintended sign (including an abnormal laboratory finding), symptom/disease temporally associated with use of investigational product, whether or not considered related to investigational product. AEs were reported based on the National Cancer Institute Common Terminology Criteria for AEs, version 4.0 (NCI-CTCAE, v4.0).
Time Frame: Baseline up to 90 days after last dose of atezolizumab (approximately 62 months)
Population: Safety-evaluable population included all randomized participants who received any amount of study treatment.
Measure: Number; unit: Percentage of participants
Arm/Group | Atezolizumab | Single Agent Chemotherapy (Vinorelbine or Gemcitabine)
Number analyzed (Participants) | 300 | 147
Percentage of participants | 91.7 | 97.3

7. Secondary Outcome: Change From Baseline in European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire - Core 30 (EORTC-QLQ-C30) Score
Description: EORTC QLQ-C30 consists of 30 questions that assess 5 aspects of patient functioning (physical, emotional, role, cognitive, and social), 3 symptom scales (fatigue, nausea and vomiting, pain), global health/quality of life, and six single items (dyspnea, insomnia, appetite loss, constipation, diarrhea, and financial difficulties). It was scored according to EORTC scoring manual (Fayers et al. 2001). All EORTC scales & single-item measures are linearly transformed so that each score has a range of 0-100. A high score for a functional/global health status scale represents a high/healthy level of functioning/HRQoL (Health-Related Quality of Life); however a high score for a symptom scale represents a high level of symptomatology or problems. A ≥10-point change in the symptoms subscale score was perceived by participants as clinically significant (Osoba et al. 1998). A positive change from baseline=improvement & negative change from baseline indicated worsening.
Time Frame: Baseline, Day 1 of each treatment cycle up to 30 days after last dose (up to approximately 55 months) (Cycle length = 21 days)
Population: ITT population included all randomized participants irrespective of whether the assigned treatment was actually received. Number analyzed is the number of participants with data available for analysis at the specified timepoint.
Measure: Mean (Standard Deviation); unit: units of a scale
Arm/Group | Atezolizumab | Single Agent Chemotherapy (Vinorelbine or Gemcitabine)
Number analyzed (Participants) | 302 | 151
units of a scale
  GHS/HRQoL Scale Score, Baseline: number analyzed (Participants) | 291 | 146
  GHS/HRQoL Scale Score, Baseline | 54.70 (22.00) | 55.25 (21.06)
  GHS/HRQoL Scale Score, Week 6: number analyzed (Participants) | 219 | 115
  GHS/HRQoL Scale Score, Week 6 | 2.09 (24.11) | 0.29 (22.94)
  GHS/HRQoL Scale Score, Week 12: number analyzed (Participants) | 148 | 63
  GHS/HRQoL Scale Score, Week 12 | 2.76 (23.42) | 1.85 (19.94)
  GHS/HRQoL Scale Score, Week 18: number analyzed (Participants) | 121 | 40
  GHS/HRQoL Scale Score, Week 18 | 4.20 (24.27) | -0.42 (19.52)
  GHS/HRQoL Scale Score, Week 24: number analyzed (Participants) | 105 | 29
  GHS/HRQoL Scale Score, Week 24 | 4.92 (23.90) | -1.72 (18.82)
  GHS/HRQoL Scale Score, Week 30: number analyzed (Participants) | 83 | 22
  GHS/HRQoL Scale Score, Week 30 | 4.32 (21.12) | 2.65 (13.70)
  GHS/HRQoL Scale Score, Week 36: number analyzed (Participants) | 62 | 16
  GHS/HRQoL Scale Score, Week 36 | 8.20 (23.55) | -0.52 (22.25)
  GHS/HRQoL Scale Score, Week 42: number analyzed (Participants) | 54 | 14
  GHS/HRQoL Scale Score, Week 42 | 6.17 (24.98) | 1.19 (19.02)
  GHS/HRQoL Scale Score, Week 48: number analyzed (Participants) | 44 | 12
  GHS/HRQoL Scale Score, Week 48 | 6.44 (27.37) | 4.86 (15.67)
  GHS/HRQoL Scale Score, Week 57: number analyzed (Participants) | 37 | 8
  GHS/HRQoL Scale Score, Week 57 | 8.56 (20.46) | 8.33 (12.60)
  GHS/HRQoL Scale Score, Week 66: number analyzed (Participants) | 33 | 5
  GHS/HRQoL Scale Score, Week 66 | 6.82 (19.15) | 5.00 (17.28)
  GHS/HRQoL Scale Score, Week 75: number analyzed (Participants) | 26 | 4
  GHS/HRQoL Scale Score, Week 75 | 3.85 (21.11) | 2.08 (24.88)
  GHS/HRQoL Scale Score, Week 84: number analyzed (Participants) | 19 | 3
  GHS/HRQoL Scale Score, Week 84 | 11.40 (20.07) | -2.78 (12.73)
  GHS/HRQoL Scale Score, Week 93: number analyzed (Participants) | 20 | 2
  GHS/HRQoL Scale Score, Week 93 | 2.08 (24.61) | -12.50 (5.89)
  GHS/HRQoL Scale Score, Week 102: number analyzed (Participants) | 16 | 1
  GHS/HRQoL Scale Score, Week 102 | 4.69 (18.50) | -25.00 (NA) — The standard deviation is a measure of the amount of variation or dispersion of a set of values. Number analyzed is 1 so standard deviation is not available.
  GHS/HRQoL Scale Score, Week 111: number analyzed (Participants) | 14 | 0
  GHS/HRQoL Scale Score, Week 111 | 1.79 (21.73) |
  GHS/HRQoL Scale Score, Week 120: number analyzed (Participants) | 14 | 0
  GHS/HRQoL Scale Score, Week 120 | 2.38 (20.52) |
  GHS/HRQoL Scale Score, Week 129: number analyzed (Participants) | 14 | 0
  GHS/HRQoL Scale Score, Week 129 | -2.98 (19.78) |
  GHS/HRQoL Scale Score, Week 138: number analyzed (Participants) | 14 | 0
  GHS/HRQoL Scale Score, Week 138 | 1.19 (25.91) |
  GHS/HRQoL Scale Score, Week 147: number analyzed (Participants) | 14 | 0
  GHS/HRQoL Scale Score, Week 147 | 4.17 (18.42) |
  GHS/HRQoL Scale Score, Week 156: number analyzed (Participants) | 7 | 0
  GHS/HRQoL Scale Score, Week 156 | -2.38 (17.82) |
  GHS/HRQoL Scale Score, Week 165: number analyzed (Participants) | 8 | 0
  GHS/HRQoL Scale Score, Week 165 | -3.13 (23.54) |
  GHS/HRQoL Scale Score, Week 174: number analyzed (Participants) | 7 | 0
  GHS/HRQoL Scale Score, Week 174 | -2.38 (17.82) |
  GHS/HRQoL Scale Score, Week 183: number analyzed (Participants) | 5 | 0
  GHS/HRQoL Scale Score, Week 183 | -6.67 (19.00) |
  GHS/HRQoL Scale Score, Week 192: number analyzed (Participants) | 4 | 0
  GHS/HRQoL Scale Score, Week 192 | -4.17 (20.97) |
  GHS/HRQoL Scale Score, Week 201: number analyzed (Participants) | 2 | 0
  GHS/HRQoL Scale Score, Week 201 | 0.00 (0.00) |
  GHS/HRQoL Scale Score, Week 210: number analyzed (Participants) | 1 | 0
  GHS/HRQoL Scale Score, Week 210 | -16.67 (NA) — The standard deviation is a measure of the amount of variation or dispersion of a set of values. Number analyzed is 1 so standard deviation is not available. |
  GHS/HRQoL Scale Score, Safety Follow-Up Visit: number analyzed (Participants) | 11 | 13
  GHS/HRQoL Scale Score, Safety Follow-Up Visit | -9.85 (24.10) | 3.85 (20.30)
  Physical Functioning, Baseline: number analyzed (Participants) | 294 | 146
  Physical Functioning, Baseline | 61.34 (25.66) | 61.97 (23.75)
  Physical Functioning, Week 6: number analyzed (Participants) | 221 | 115
  Physical Functioning, Week 6 | -2.93 (17.69) | -1.07 (18.49)
  Physical Functioning, Week 12: number analyzed (Participants) | 149 | 64
  Physical Functioning, Week 12 | 0.17 (20.35) | 1.46 (18.07)
  Physical Functioning, Week 18: number analyzed (Participants) | 121 | 39
  Physical Functioning, Week 18 | 3.02 (17.97) | -1.58 (18.00)
  Physical Functioning, Week 24: number analyzed (Participants) | 107 | 30
  Physical Functioning, Week 24 | 3.49 (18.66) | -5.50 (15.64)
  Physical Functioning, Week 30: number analyzed (Participants) | 84 | 23
  Physical Functioning, Week 30 | 4.25 (18.22) | -1.23 (21.80)
  Physical Functioning, Week 36: number analyzed (Participants) | 63 | 16
  Physical Functioning, Week 36 | 6.98 (19.68) | -4.90 (28.33)
  Physical Functioning, Week 42: number analyzed (Participants) | 54 | 14
  Physical Functioning, Week 42 | 3.58 (24.08) | 0.95 (16.92)
  Physical Functioning, Week 48: number analyzed (Participants) | 43 | 12
  Physical Functioning, Week 48 | 7.44 (18.92) | 2.22 (19.76)
  Physical Functioning, Week 57: number analyzed (Participants) | 36 | 8
  Physical Functioning, Week 57 | 7.59 (16.73) | -3.33 (20.47)
  Physical Functioning, Week 66: number analyzed (Participants) | 33 | 5
  Physical Functioning, Week 66 | 4.65 (22.39) | 2.67 (17.38)
  Physical Functioning, Week 75: number analyzed (Participants) | 26 | 4
  Physical Functioning, Week 75 | 4.87 (27.88) | -1.67 (34.16)
  Physical Functioning, Week 84: number analyzed (Participants) | 18 | 3
  Physical Functioning, Week 84 | 3.70 (23.68) | -8.89 (26.94)
  Physical Functioning, Week 93: number analyzed (Participants) | 20 | 2
  Physical Functioning, Week 93 | 1.67 (23.38) | -26.67 (18.86)
  Physical Functioning, Week 102: number analyzed (Participants) | 16 | 1
  Physical Functioning, Week 102 | 2.40 (16.19) | -40.00 (NA) — The standard deviation is a measure of the amount of variation or dispersion of a set of values. Number analyzed is 1 so standard deviation is not available.
  Physical Functioning, Week 111: number analyzed (Participants) | 14 | 0
  Physical Functioning, Week 111 | 2.38 (19.67) |
  Physical Functioning, Week 120: number analyzed (Participants) | 14 | 0
  Physical Functioning, Week 120 | 3.33 (20.04) |
  Physical Functioning, Week 129: number analyzed (Participants) | 13 | 0
  Physical Functioning, Week 129 | -1.03 (19.02) |
  Physical Functioning, Week 138: number analyzed (Participants) | 14 | 0
  Physical Functioning, Week 138 | -0.48 (19.47) |
  Physical Functioning, Week 147: number analyzed (Participants) | 14 | 0
  Physical Functioning, Week 147 | -0.48 (17.04) |
  Physical Functioning, Week 156: number analyzed (Participants) | 7 | 0
  Physical Functioning, Week 156 | -4.76 (10.69) |
  Physical Functioning, Week 165: number analyzed (Participants) | 8 | 0
  Physical Functioning, Week 165 | -3.61 (13.44) |
  Physical Functioning, Week 174: number analyzed (Participants) | 7 | 0
  Physical Functioning, Week 174 | -1.90 (21.33) |
  Physical Functioning, Week 183: number analyzed (Participants) | 5 | 0
  Physical Functioning, Week 183 | 2.67 (19.21) |
  Physical Functioning, Week 192: number analyzed (Participants) | 4 | 0
  Physical Functioning, Week 192 | -3.33 (12.77) |
  Physical Functioning, Week 201: number analyzed (Participants) | 2 | 0
  Physical Functioning, Week 201 | -3.33 (4.71) |
  Physical Functioning, Week 210: number analyzed (Participants) | 1 | 0
  Physical Functioning, Week 210 | -20.00 (NA) — The standard deviation is a measure of the amount of variation or dispersion of a set of values. Number analyzed is 1 so standard deviation is not available. |
  Physical Functioning, Safety Follow-Up Visit: number analyzed (Participants) | 11 | 13
  Physical Functioning, Safety Follow-Up Visit | -9.70 (25.01) | -6.67 (27.08)
  Role Functioning, Baseline: number analyzed (Participants) | 294 | 145
  Role Functioning, Baseline | 62.53 (33.17) | 61.72 (34.31)
  Role Functioning, Week 6: number analyzed (Participants) | 222 | 114
  Role Functioning, Week 6 | -2.63 (28.13) | -3.51 (30.12)
  Role Functioning, Week 12: number analyzed (Participants) | 150 | 63
  Role Functioning, Week 12 | -1.78 (30.48) | -1.59 (26.56)
  Role Functioning, Week 18: number analyzed (Participants) | 122 | 39
  Role Functioning, Week 18 | -0.96 (30.02) | 1.71 (36.63)
  Role Functioning, Week 24: number analyzed (Participants) | 107 | 30
  Role Functioning, Week 24 | 1.25 (30.00) | -5.00 (28.42)
  Role Functioning, Week 30: number analyzed (Participants) | 84 | 23
  Role Functioning, Week 30 | -0.20 (29.10) | -7.25 (32.50)
  Role Functioning, Week 36: number analyzed (Participants) | 62 | 16
  Role Functioning, Week 36 | 2.15 (35.00) | -14.58 (47.09)
  Role Functioning, Week 42: number analyzed (Participants) | 54 | 14
  Role Functioning, Week 42 | 1.54 (35.95) | -4.76 (47.78)
  Role Functioning, Week 48: number analyzed (Participants) | 44 | 12
  Role Functioning, Week 48 | 4.92 (29.55) | -2.78 (34.69)
  Role Functioning, Week 57: number analyzed (Participants) | 37 | 8
  Role Functioning, Week 57 | 3.15 (28.82) | -4.17 (19.42)
  Role Functioning, Week 66: number analyzed (Participants) | 33 | 5
  Role Functioning, Week 66 | 0.51 (25.17) | -6.67 (25.28)
  Role Functioning, Week 75: number analyzed (Participants) | 26 | 4
  Role Functioning, Week 75 | -0.64 (31.44) | 8.33 (48.11)
  Role Functioning, Week 84: number analyzed (Participants) | 18 | 3
  Role Functioning, Week 84 | 3.70 (16.72) | -11.11 (19.25)
  Role Functioning, Week 93: number analyzed (Participants) | 20 | 2
  Role Functioning, Week 93 | -1.67 (26.98) | -25.00 (35.36)
  Role Functioning, Week 102: number analyzed (Participants) | 16 | 1
  Role Functioning, Week 102 | 2.08 (18.13) | -33.33 (NA) — The standard deviation is a measure of the amount of variation or dispersion of a set of values. Number analyzed is 1 so standard deviation is not available.
  Role Functioning, Week 111: number analyzed (Participants) | 14 | 0
  Role Functioning, Week 111 | -3.57 (22.81) |
  Role Functioning, Week 120: number analyzed (Participants) | 14 | 0
  Role Functioning, Week 120 | -1.19 (19.02) |
  Role Functioning, Week 129: number analyzed (Participants) | 14 | 0
  Role Functioning, Week 129 | -1.19 (17.86) |
  Role Functioning, Week 138: number analyzed (Participants) | 14 | 0
  Role Functioning, Week 138 | -2.38 (22.51) |
  Role Functioning, Week 147: number analyzed (Participants) | 14 | 0
  Role Functioning, Week 147 | -3.57 (17.52) |
  Role Functioning, Week 156: number analyzed (Participants) | 7 | 0
  Role Functioning, Week 156 | -2.38 (6.30) |
  Role Functioning, Week 165: number analyzed (Participants) | 8 | 0
  Role Functioning, Week 165 | -10.42 (26.63) |
  Role Functioning, Week 174: number analyzed (Participants) | 7 | 0
  Role Functioning, Week 174 | -7.14 (26.97) |
  Role Functioning, Week 183: number analyzed (Participants) | 5 | 0
  Role Functioning, Week 183 | -10.00 (9.13) |
  Role Functioning, Week 192: number analyzed (Participants) | 4 | 0
  Role Functioning, Week 192 | -16.67 (13.61) |
  Role Functioning, Week 201: number analyzed (Participants) | 2 | 0
  Role Functioning, Week 201 | 0.00 (0.00) |
  Role Functioning, Week 210: number analyzed (Participants) | 1 | 0
  Role Functioning, Week 210 | 0.00 (NA) — The standard deviation is a measure of the amount of variation or dispersion of a set of values. Number analyzed is 1 so standard deviation is not available. |
  Role Functioning, Safety Follow-Up Visit: number analyzed (Participants) | 11 | 13
  Role Functioning, Safety Follow-Up Visit | -22.73 (41.01) | -1.28 (43.28)
  Emotional Functioning, Baseline: number analyzed (Participants) | 290 | 146
  Emotional Functioning, Baseline | 74.20 (23.87) | 73.38 (23.55)
  Emotional Functioning, Week 6: number analyzed (Participants) | 219 | 115
  Emotional Functioning, Week 6 | 2.12 (20.59) | 0.46 (23.00)
  Emotional Functioning, Week 12: number analyzed (Participants) | 148 | 64
  Emotional Functioning, Week 12 | 1.24 (21.06) | 4.21 (22.77)
  Emotional Functioning, Week 18: number analyzed (Participants) | 120 | 40
  Emotional Functioning, Week 18 | 3.82 (18.23) | 0.28 (22.10)
  Emotional Functioning, Week 24: number analyzed (Participants) | 105 | 30
  Emotional Functioning, Week 24 | 4.13 (17.07) | 4.07 (17.40)
  Emotional Functioning, Week 30: number analyzed (Participants) | 83 | 23
  Emotional Functioning, Week 30 | 3.15 (17.62) | 2.17 (20.29)
  Emotional Functioning, Week 36: number analyzed (Participants) | 62 | 16
  Emotional Functioning, Week 36 | 2.02 (16.78) | -5.38 (21.31)
  Emotional Functioning, Week 42: number analyzed (Participants) | 54 | 14
  Emotional Functioning, Week 42 | 2.01 (19.08) | -7.14 (16.30)
  Emotional Functioning, Week 48: number analyzed (Participants) | 43 | 12
  Emotional Functioning, Week 48 | 5.04 (13.87) | -3.47 (10.33)
  Emotional Functioning, Week 57: number analyzed (Participants) | 37 | 8
  Emotional Functioning, Week 57 | 5.78 (20.58) | 3.13 (23.12)
  Emotional Functioning, Week 66: number analyzed (Participants) | 33 | 5
  Emotional Functioning, Week 66 | 4.29 (17.81) | 6.67 (6.97)
  Emotional Functioning, Week 75: number analyzed (Participants) | 26 | 4
  Emotional Functioning, Week 75 | 0.32 (21.01) | 12.50 (28.46)
  Emotional Functioning, Week 84: number analyzed (Participants) | 19 | 3
  Emotional Functioning, Week 84 | 6.58 (17.91) | 0.00 (16.97)
  Emotional Functioning, Week 93: number analyzed (Participants) | 20 | 2
  Emotional Functioning, Week 93 | 2.92 (13.59) | -4.17 (5.89)
  Emotional Functioning, Week 102: number analyzed (Participants) | 16 | 1
  Emotional Functioning, Week 102 | 4.69 (12.53) | -16.67 (NA) — The standard deviation is a measure of the amount of variation or dispersion of a set of values. Number analyzed is 1 so standard deviation is not available.
  Emotional Functioning, Week 111: number analyzed (Participants) | 14 | 0
  Emotional Functioning, Week 111 | 3.57 (15.92) |
  Emotional Functioning, Week 120: number analyzed (Participants) | 14 | 0
  Emotional Functioning, Week 120 | 1.79 (10.93) |
  Emotional Functioning, Week 129: number analyzed (Participants) | 14 | 0
  Emotional Functioning, Week 129 | 2.98 (12.91) |
  Emotional Functioning, Week 138: number analyzed (Participants) | 14 | 0
  Emotional Functioning, Week 138 | 4.17 (12.97) |
  Emotional Functioning, Week 147: number analyzed (Participants) | 14 | 0
  Emotional Functioning, Week 147 | 5.36 (18.08) |
  Emotional Functioning, Week 156: number analyzed (Participants) | 7 | 0
  Emotional Functioning, Week 156 | 2.38 (10.45) |
  Emotional Functioning, Week 165: number analyzed (Participants) | 8 | 0
  Emotional Functioning, Week 165 | -1.04 (8.26) |
  Emotional Functioning, Week 174: number analyzed (Participants) | 7 | 0
  Emotional Functioning, Week 174 | 2.38 (12.47) |
  Emotional Functioning, Week 183: number analyzed (Participants) | 5 | 0
  Emotional Functioning, Week 183 | -1.67 (10.87) |
  Emotional Functioning, Week 192: number analyzed (Participants) | 4 | 0
  Emotional Functioning, Week 192 | -2.08 (10.49) |
  Emotional Functioning, Week 201: number analyzed (Participants) | 2 | 0
  Emotional Functioning, Week 201 | -4.17 (17.68) |
  Emotional Functioning, Week 210: number analyzed (Participants) | 1 | 0
  Emotional Functioning, Week 210 | -16.67 (NA) — The standard deviation is a measure of the amount of variation or dispersion of a set of values. Number analyzed is 1 so standard deviation is not available. |
  Emotional Functioning, Safety Follow-Up Visit: number analyzed (Participants) | 11 | 13
  Emotional Functioning, Safety Follow-Up Visit | 6.82 (26.57) | -5.77 (21.08)
  Cognitive Functioning, Baseline: number analyzed (Participants) | 291 | 146
  Cognitive Functioning, Baseline | 81.39 (21.49) | 82.65 (19.95)
  Cognitive Functioning, Week 6: number analyzed (Participants) | 219 | 115
  Cognitive Functioning, Week 6 | -1.67 (21.17) | -5.94 (21.76)
  Cognitive Functioning, Week 12: number analyzed (Participants) | 149 | 64
  Cognitive Functioning, Week 12 | -1.79 (22.52) | -2.60 (22.27)
  Cognitive Functioning, Week 18: number analyzed (Participants) | 121 | 40
  Cognitive Functioning, Week 18 | 2.62 (19.95) | -7.92 (24.46)
  Cognitive Functioning, Week 24: number analyzed (Participants) | 105 | 30
  Cognitive Functioning, Week 24 | 0.48 (18.41) | -10.00 (28.57)
  Cognitive Functioning, Week 30: number analyzed (Participants) | 83 | 23
  Cognitive Functioning, Week 30 | -2.01 (18.11) | -8.70 (17.31)
  Cognitive Functioning, Week 36: number analyzed (Participants) | 62 | 16
  Cognitive Functioning, Week 36 | -0.54 (15.96) | -11.46 (16.91)
  Cognitive Functioning, Week 42: number analyzed (Participants) | 54 | 14
  Cognitive Functioning, Week 42 | -4.94 (23.71) | -7.14 (12.60)
  Cognitive Functioning, Week 48: number analyzed (Participants) | 44 | 12
  Cognitive Functioning, Week 48 | -1.89 (16.16) | -11.11 (14.79)
  Cognitive Functioning, Week 57: number analyzed (Participants) | 37 | 8
  Cognitive Functioning, Week 57 | -3.15 (20.73) | -2.08 (16.52)
  Cognitive Functioning, Week 66: number analyzed (Participants) | 33 | 5
  Cognitive Functioning, Week 66 | -4.04 (23.58) | -3.33 (18.26)
  Cognitive Functioning, Week 75: number analyzed (Participants) | 26 | 4
  Cognitive Functioning, Week 75 | -5.13 (17.49) | -4.17 (20.97)
  Cognitive Functioning, Week 84: number analyzed (Participants) | 19 | 3
  Cognitive Functioning, Week 84 | -3.51 (18.90) | 5.56 (9.62)
  Cognitive Functioning, Week 93: number analyzed (Participants) | 20 | 2
  Cognitive Functioning, Week 93 | 3.33 (12.80) | 0.00 (0.00)
  Cognitive Functioning, Week 102: number analyzed (Participants) | 16 | 1
  Cognitive Functioning, Week 102 | 4.17 (16.67) | 0.00 (NA) — The standard deviation is a measure of the amount of variation or dispersion of a set of values. Number analyzed is 1 so standard deviation is not available.
  Cognitive Functioning, Week 111: number analyzed (Participants) | 14 | 0
  Cognitive Functioning, Week 111 | 4.76 (16.57) |
  Cognitive Functioning, Week 120: number analyzed (Participants) | 14 | 0
  Cognitive Functioning, Week 120 | 0.00 (20.67) |
  Cognitive Functioning, Week 129: number analyzed (Participants) | 14 | 0
  Cognitive Functioning, Week 129 | 0.00 (13.07) |
  Cognitive Functioning, Week 138: number analyzed (Participants) | 14 | 0
  Cognitive Functioning, Week 138 | -2.38 (20.52) |
  Cognitive Functioning, Week 147: number analyzed (Participants) | 14 | 0
  Cognitive Functioning, Week 147 | 1.19 (16.62) |
  Cognitive Functioning, Week 156: number analyzed (Participants) | 7 | 0
  Cognitive Functioning, Week 156 | 4.76 (12.60) |
  Cognitive Functioning, Week 165: number analyzed (Participants) | 8 | 0
  Cognitive Functioning, Week 165 | 6.25 (12.40) |
  Cognitive Functioning, Week 174: number analyzed (Participants) | 7 | 0
  Cognitive Functioning, Week 174 | 0.00 (9.62) |
  Cognitive Functioning, Week 183: number analyzed (Participants) | 5 | 0
  Cognitive Functioning, Week 183 | 3.33 (18.26) |
  Cognitive Functioning, Week 192: number analyzed (Participants) | 4 | 0
  Cognitive Functioning, Week 192 | 0.00 (0.00) |
  Cognitive Functioning, Week 201: number analyzed (Participants) | 2 | 0
  Cognitive Functioning, Week 201 | 0.00 (0.00) |
  Cognitive Functioning, Week 210: number analyzed (Participants) | 1 | 0
  Cognitive Functioning, Week 210 | 0.00 (NA) — The standard deviation is a measure of the amount of variation or dispersion of a set of values. Number analyzed is 1 so standard deviation is not available. |
  Cognitive Functioning, Safety Follow-Up Visit: number analyzed (Participants) | 11 | 13
  Cognitive Functioning, Safety Follow-Up Visit | -16.67 (23.57) | 5.13 (25.81)
  Social Functioning, Baseline: number analyzed (Participants) | 290 | 146
  Social Functioning, Baseline | 71.32 (29.12) | 74.43 (27.62)
  Social Functioning, Week 6: number analyzed (Participants) | 218 | 115
  Social Functioning, Week 6 | 1.30 (27.66) | -4.49 (28.30)
  Social Functioning, Week 12: number analyzed (Participants) | 148 | 64
  Social Functioning, Week 12 | 1.58 (27.93) | -4.17 (32.93)
  Social Functioning, Week 18: number analyzed (Participants) | 119 | 40
  Social Functioning, Week 18 | 5.60 (24.38) | -14.17 (31.93)
  Social Functioning, Week 24: number analyzed (Participants) | 105 | 30
  Social Functioning, Week 24 | 5.08 (24.91) | -11.11 (27.45)
  Social Functioning, Week 30: number analyzed (Participants) | 83 | 23
  Social Functioning, Week 30 | 4.82 (23.79) | -5.80 (36.10)
  Social Functioning, Week 36: number analyzed (Participants) | 61 | 16
  Social Functioning, Week 36 | 3.01 (27.97) | -14.58 (42.11)
  Social Functioning, Week 42: number analyzed (Participants) | 54 | 14
  Social Functioning, Week 42 | -0.31 (26.79) | -7.14 (36.23)
  Social Functioning, Week 48: number analyzed (Participants) | 44 | 12
  Social Functioning, Week 48 | 1.89 (21.93) | -5.56 (28.72)
  Social Functioning, Week 57: number analyzed (Participants) | 37 | 8
  Social Functioning, Week 57 | 3.60 (29.17) | 2.08 (30.13)
  Social Functioning, Week 66: number analyzed (Participants) | 33 | 5
  Social Functioning, Week 66 | 5.56 (26.90) | 3.33 (29.81)
  Social Functioning, Week 75: number analyzed (Participants) | 26 | 4
  Social Functioning, Week 75 | 5.77 (23.07) | 4.17 (34.36)
  Social Functioning, Week 84: number analyzed (Participants) | 19 | 3
  Social Functioning, Week 84 | 2.63 (21.70) | 22.22 (25.46)
  Social Functioning, Week 93: number analyzed (Participants) | 20 | 2
  Social Functioning, Week 93 | 8.33 (16.67) | 8.33 (11.79)
  Social Functioning, Week 102: number analyzed (Participants) | 16 | 1
  Social Functioning, Week 102 | 9.38 (17.18) | 16.67 (NA) — The standard deviation is a measure of the amount of variation or dispersion of a set of values. Number analyzed is 1 so standard deviation is not available.
  Social Functioning, Week 111: number analyzed (Participants) | 14 | 0
  Social Functioning, Week 111 | 2.38 (18.32) |
  Social Functioning, Week 120: number analyzed (Participants) | 14 | 0
  Social Functioning, Week 120 | 7.14 (14.19) |
  Social Functioning, Week 129: number analyzed (Participants) | 14 | 0
  Social Functioning, Week 129 | -2.38 (30.56) |
  Social Functioning, Week 138: number analyzed (Participants) | 14 | 0
  Social Functioning, Week 138 | 2.38 (20.52) |
  Social Functioning, Week 147: number analyzed (Participants) | 14 | 0
  Social Functioning, Week 147 | 7.14 (16.94) |
  Social Functioning, Week 156: number analyzed (Participants) | 7 | 0
  Social Functioning, Week 156 | 4.76 (15.85) |
  Social Functioning, Week 165: number analyzed (Participants) | 8 | 0
  Social Functioning, Week 165 | -6.25 (29.46) |
  Social Functioning, Week 174: number analyzed (Participants) | 7 | 0
  Social Functioning, Week 174 | 7.14 (26.97) |
  Social Functioning, Week 183: number analyzed (Participants) | 5 | 0
  Social Functioning, Week 183 | 6.67 (38.37) |
  Social Functioning, Week 192: number analyzed (Participants) | 4 | 0
  Social Functioning, Week 192 | -4.17 (28.46) |
  Social Functioning, Week 201: number analyzed (Participants) | 2 | 0
  Social Functioning, Week 201 | -25.00 (35.36) |
  Social Functioning, Week 210: number analyzed (Participants) | 1 | 0
  Social Functioning, Week 210 | -50.00 (NA) — The standard deviation is a measure of the amount of variation or dispersion of a set of values. Number analyzed is 1 so standard deviation is not available. |
  Social Functioning, Safety Follow-Up Visit: number analyzed (Participants) | 11 | 13
  Social Functioning, Safety Follow-Up Visit | 1.52 (46.22) | -12.82 (34.80)
  Fatigue, Baseline: number analyzed (Participants) | 293 | 146
  Fatigue, Baseline | 41.62 (26.98) | 42.62 (25.10)
  Fatigue, Week 6: number analyzed (Participants) | 221 | 115
  Fatigue, Week 6 | 3.37 (23.32) | 2.08 (23.71)
  Fatigue, Week 12: number analyzed (Participants) | 148 | 64
  Fatigue, Week 12 | 0.53 (26.98) | -1.56 (22.99)
  Fatigue, Week 18: number analyzed (Participants) | 121 | 40
  Fatigue, Week 18 | -1.79 (22.11) | 2.22 (18.69)
  Fatigue, Week 24: number analyzed (Participants) | 106 | 30
  Fatigue, Week 24 | -3.14 (25.82) | 2.96 (21.43)
  Fatigue, Week 30: number analyzed (Participants) | 83 | 23
  Fatigue, Week 30 | -2.88 (22.98) | -3.38 (24.03)
  Fatigue, Week 36: number analyzed (Participants) | 63 | 16
  Fatigue, Week 36 | -4.06 (28.12) | 4.86 (27.81)
  Fatigue, Week 42: number analyzed (Participants) | 54 | 14
  Fatigue, Week 42 | -2.67 (29.11) | 3.17 (28.05)
  Fatigue, Week 48: number analyzed (Participants) | 43 | 12
  Fatigue, Week 48 | -6.72 (24.86) | 1.85 (23.61)
  Fatigue, Week 57: number analyzed (Participants) | 37 | 8
  Fatigue, Week 57 | -3.30 (22.66) | 1.39 (18.25)
  Fatigue, Week 66: number analyzed (Participants) | 33 | 5
  Fatigue, Week 66 | -2.53 (29.63) | -6.67 (12.67)
  Fatigue, Week 75: number analyzed (Participants) | 26 | 4
  Fatigue, Week 75 | -4.70 (22.26) | -8.33 (33.18)
  Fatigue, Week 84: number analyzed (Participants) | 18 | 3
  Fatigue, Week 84 | -6.79 (26.72) | 22.22 (19.25)
  Fatigue, Week 93: number analyzed (Participants) | 20 | 2
  Fatigue, Week 93 | -5.56 (30.05) | 22.22 (0.00)
  Fatigue, Week 102: number analyzed (Participants) | 16 | 1
  Fatigue, Week 102 | -5.56 (26.91) | 33.33 (NA) — The standard deviation is a measure of the amount of variation or dispersion of a set of values. Number analyzed is 1 so standard deviation is not available.
  Fatigue, Week 111: number analyzed (Participants) | 14 | 0
  Fatigue, Week 111 | -0.79 (33.32) |
  Fatigue, Week 120: number analyzed (Participants) | 14 | 0
  Fatigue, Week 120 | -2.38 (28.30) |
  Fatigue, Week 129: number analyzed (Participants) | 14 | 0
  Fatigue, Week 129 | -2.78 (18.33) |
  Fatigue, Week 138: number analyzed (Participants) | 14 | 0
  Fatigue, Week 138 | -1.59 (26.10) |
  Fatigue, Week 147: number analyzed (Participants) | 14 | 0
  Fatigue, Week 147 | -3.17 (25.94) |
  Fatigue, Week 156: number analyzed (Participants) | 7 | 0
  Fatigue, Week 156 | -1.59 (14.95) |
  Fatigue, Week 165: number analyzed (Participants) | 8 | 0
  Fatigue, Week 165 | 1.39 (29.95) |
  Fatigue, Week 174: number analyzed (Participants) | 7 | 0
  Fatigue, Week 174 | -4.76 (20.14) |
  Fatigue, Week 183: number analyzed (Participants) | 5 | 0
  Fatigue, Week 183 | 4.44 (26.76) |
  Fatigue, Week 192: number analyzed (Participants) | 4 | 0
  Fatigue, Week 192 | 5.56 (14.34) |
  Fatigue, Week 201: number analyzed (Participants) | 2 | 0
  Fatigue, Week 201 | -5.56 (7.86) |
  Fatigue, Week 210: number analyzed (Participants) | 1 | 0
  Fatigue, Week 210 | -11.11 (NA) — The standard deviation is a measure of the amount of variation or dispersion of a set of values. Number analyzed is 1 so standard deviation is not available. |
  Fatigue, Safety Follow-Up Visit: number analyzed (Participants) | 11 | 13
  Fatigue, Safety Follow-Up Visit | 0.00 (31.82) | 1.71 (33.59)
  Nausea and Vomiting, Baseline: number analyzed (Participants) | 294 | 146
  Nausea and Vomiting, Baseline | 8.28 (17.07) | 7.99 (15.06)
  Nausea and Vomiting, Week 6: number analyzed (Participants) | 222 | 115
  Nausea and Vomiting, Week 6 | 0.90 (16.98) | 1.01 (19.28)
  Nausea and Vomiting, Week 12: number analyzed (Participants) | 149 | 64
  Nausea and Vomiting, Week 12 | 1.12 (17.72) | 3.65 (16.92)
  Nausea and Vomiting, Week 18: number analyzed (Participants) | 122 | 40
  Nausea and Vomiting, Week 18 | -0.41 (15.67) | 3.33 (18.18)
  Nausea and Vomiting, Week 24: number analyzed (Participants) | 107 | 30
  Nausea and Vomiting, Week 24 | -1.87 (14.54) | 3.33 (16.02)
  Nausea and Vomiting, Week 30: number analyzed (Participants) | 84 | 23
  Nausea and Vomiting, Week 30 | -2.38 (16.39) | 3.62 (10.0063)
  Nausea and Vomiting, Week 36: number analyzed (Participants) | 63 | 16
  Nausea and Vomiting, Week 36 | 2.12 (17.32) | 3.13 (15.18)
  Nausea and Vomiting, Week 42: number analyzed (Participants) | 54 | 14
  Nausea and Vomiting, Week 42 | 1.54 (11.79) | 3.57 (19.81)
  Nausea and Vomiting, Week 48: number analyzed (Participants) | 43 | 12
  Nausea and Vomiting, Week 48 | -1.55 (15.78) | 0.00 (20.10)
  Nausea and Vomiting, Week 57: number analyzed (Participants) | 37 | 8
  Nausea and Vomiting, Week 57 | 2.25 (11.89) | 2.08 (18.77)
  Nausea and Vomiting, Week 66: number analyzed (Participants) | 33 | 5
  Nausea and Vomiting, Week 66 | -1.01 (14.99) | -3.33 (7.45)
  Nausea and Vomiting, Week 75: number analyzed (Participants) | 26 | 4
  Nausea and Vomiting, Week 75 | 2.56 (9.06) | -4.17 (8.33)
  Nausea and Vomiting, Week 84: number analyzed (Participants) | 19 | 3
  Nausea and Vomiting, Week 84 | 0.88 (8.74) | 0.00 (16.67)
  Nausea and Vomiting, Week 93: number analyzed (Participants) | 20 | 2
  Nausea and Vomiting, Week 93 | -1.67 (5.13) | -8.33 (11.79)
  Nausea and Vomiting, Week 102: number analyzed (Participants) | 16 | 1
  Nausea and Vomiting, Week 102 | -2.08 (5.69) | 0.00 (NA) — The standard deviation is a measure of the amount of variation or dispersion of a set of values. Number analyzed is 1 so standard deviation is not available.
  Nausea and Vomiting, Week 111: number analyzed (Participants) | 14 | 0
  Nausea and Vomiting, Week 111 | 4.76 (12.10) |
  Nausea and Vomiting, Week 120: number analyzed (Participants) | 14 | 0
  Nausea and Vomiting, Week 120 | -1.19 (7.91) |
  Nausea and Vomiting, Week 129: number analyzed (Participants) | 14 | 0
  Nausea and Vomiting, Week 129 | 0.00 (6.54) |
  Nausea and Vomiting, Week 138: number analyzed (Participants) | 14 | 0
  Nausea and Vomiting, Week 138 | -2.38 (6.05) |
  Nausea and Vomiting, Week 147: number analyzed (Participants) | 14 | 0
  Nausea and Vomiting, Week 147 | -2.38 (6.05) |
  Nausea and Vomiting, Week 156: number analyzed (Participants) | 7 | 0
  Nausea and Vomiting, Week 156 | -2.38 (6.30) |
  Nausea and Vomiting, Week 165: number analyzed (Participants) | 8 | 0
  Nausea and Vomiting, Week 165 | -2.08 (5.89) |
  Nausea and Vomiting, Week 174: number analyzed (Participants) | 7 | 0
  Nausea and Vomiting, Week 174 | -2.38 (6.30) |
  Nausea and Vomiting, Week 183: number analyzed (Participants) | 5 | 0
  Nausea and Vomiting, Week 183 | -3.33 (7.45) |
  Nausea and Vomiting, Week 192: number analyzed (Participants) | 4 | 0
  Nausea and Vomiting, Week 192 | 0.00 (0.00) |
  Nausea and Vomiting, Week 201: number analyzed (Participants) | 2 | 0
  Nausea and Vomiting, Week 201 | 0.00 (0.00) |
  Nausea and Vomiting, Week 210: number analyzed (Participants) | 1 | 0
  Nausea and Vomiting, Week 210 | 0.00 (NA) — The standard deviation is a measure of the amount of variation or dispersion of a set of values. Number analyzed is 1 so standard deviation is not available. |
  Nausea and Vomiting, Safety Follow-Up Visit: number analyzed (Participants) | 11 | 13
  Nausea and Vomiting, Safety Follow-Up Visit | 13.64 (42.04) | 0.00 (33.33)
  Pain, Baseline: number analyzed (Participants) | 294 | 146
  Pain, Baseline | 31.52 (29.67) | 32.99 (29.06)
  Pain, Week 6: number analyzed (Participants) | 222 | 115
  Pain, Week 6 | -0.98 (25.27) | -1.01 (26.61)
  Pain, Week 12: number analyzed (Participants) | 149 | 64
  Pain, Week 12 | -3.58 (29.67) | -5.73 (27.09)
  Pain, Week 18: number analyzed (Participants) | 121 | 40
  Pain, Week 18 | -5.51 (30.38) | 3.75 (31.23)
  Pain, Week 24: number analyzed (Participants) | 107 | 30
  Pain, Week 24 | -6.70 (30.01) | 3.89 (23.44)
  Pain, Week 30: number analyzed (Participants) | 84 | 23
  Pain, Week 30 | -5.36 (30.30) | -9.42 (21.80)
  Pain, Week 36: number analyzed (Participants) | 63 | 16
  Pain, Week 36 | -7.41 (28.36) | 3.13 (25.25)
  Pain, Week 42: number analyzed (Participants) | 54 | 14
  Pain, Week 42 | -5.25 (33.77) | -4.76 (33.61)
  Pain, Week 48: number analyzed (Participants) | 44 | 12
  Pain, Week 48 | -9.85 (30.57) | -11.11 (26.91)
  Pain, Week 57: number analyzed (Participants) | 37 | 8
  Pain, Week 57 | -7.21 (31.80) | -6.25 (25.10)
  Pain, Week 66: number analyzed (Participants) | 33 | 5
  Pain, Week 66 | -13.13 (30.26) | -20.00 (21.73)
  Pain, Week 75: number analyzed (Participants) | 26 | 4
  Pain, Week 75 | -5.77 (33.65) | 0.00 (36.00)
  Pain, Week 84: number analyzed (Participants) | 19 | 3
  Pain, Week 84 | -15.79 (26.34) | -11.11 (19.25)
  Pain, Week 93: number analyzed (Participants) | 20 | 2
  Pain, Week 93 | -7.50 (27.29) | -16.67 (23.57)
  Pain, Week 102: number analyzed (Participants) | 16 | 1
  Pain, Week 102 | -17.71 (25.44) | -33.33 (NA) — The standard deviation is a measure of the amount of variation or dispersion of a set of values. Number analyzed is 1 so standard deviation is not available.
  Pain, Week 111: number analyzed (Participants) | 14 | 0
  Pain, Week 111 | -14.29 (23.44) |
  Pain, Week 120: number analyzed (Participants) | 14 | 0
  Pain, Week 120 | -15.48 (26.53) |
  Pain, Week 129: number analyzed (Participants) | 14 | 0
  Pain, Week 129 | -10.71 (16.80) |
  Pain, Week 138: number analyzed (Participants) | 14 | 0
  Pain, Week 138 | -15.48 (25.71) |
  Pain, Week 147: number analyzed (Participants) | 14 | 0
  Pain, Week 147 | -13.10 (27.87) |
  Pain, Week 156: number analyzed (Participants) | 7 | 0
  Pain, Week 156 | -14.29 (20.25) |
  Pain, Week 165: number analyzed (Participants) | 8 | 0
  Pain, Week 165 | -10.42 (19.80) |
  Pain, Week 174: number analyzed (Participants) | 7 | 0
  Pain, Week 174 | -11.90 (34.31) |
  Pain, Week 183: number analyzed (Participants) | 5 | 0
  Pain, Week 183 | -13.33 (36.13) |
  Pain, Week 192: number analyzed (Participants) | 4 | 0
  Pain, Week 192 | -12.50 (25.00) |
  Pain, Week 201: number analyzed (Participants) | 2 | 0
  Pain, Week 201 | -25.00 (35.36) |
  Pain, Week 210: number analyzed (Participants) | 1 | 0
  Pain, Week 210 | -16.67 (NA) — The standard deviation is a measure of the amount of variation or dispersion of a set of values. Number analyzed is 1 so standard deviation is not available. |
  Pain, Safety Follow-Up Visit: number analyzed (Participants) | 11 | 13
  Pain, Safety Follow-Up Visit | 9.09 (26.21) | -7.69 (38.26)
  Dyspnoea, Baseline: number analyzed (Participants) | 294 | 145
  Dyspnoea, Baseline | 36.17 (30.47) | 39.31 (31.35)
  Dyspnoea, Week 6: number analyzed (Participants) | 220 | 114
  Dyspnoea, Week 6 | -1.36 (28.55) | -0.58 (29.74)
  Dyspnoea, Week 12: number analyzed (Participants) | 149 | 64
  Dyspnoea, Week 12 | 0.45 (30.51) | -4.69 (27.13)
  Dyspnoea, Week 18: number analyzed (Participants) | 122 | 40
  Dyspnoea, Week 18 | -1.91 (26.87) | -3.33 (31.85)
  Dyspnoea, Week 24: number analyzed (Participants) | 106 | 30
  Dyspnoea, Week 24 | -5.03 (29.02) | -4.44 (29.99)
  Dyspnoea, Week 30: number analyzed (Participants) | 84 | 23
  Dyspnoea, Week 30 | -4.37 (28.24) | -8.70 (30.51)
  Dyspnoea, Week 36: number analyzed (Participants) | 62 | 16
  Dyspnoea, Week 36 | -6.99 (27.08) | 0.00 (34.43)
  Dyspnoea, Week 42: number analyzed (Participants) | 54 | 13
  Dyspnoea, Week 42 | -8.64 (32.50) | -7.69 (19.97)
  Dyspnoea, Week 48: number analyzed (Participants) | 44 | 11
  Dyspnoea, Week 48 | -7.58 (30.38) | -3.03 (23.35)
  Dyspnoea, Week 57: number analyzed (Participants) | 37 | 8
  Dyspnoea, Week 57 | -9.01 (30.07) | -12.50 (24.80)
  Dyspnoea, Week 66: number analyzed (Participants) | 33 | 5
  Dyspnoea, Week 66 | -3.03 (30.46) | -20.00 (18.26)
  Dyspnoea, Week 75: number analyzed (Participants) | 26 | 4
  Dyspnoea, Week 75 | -5.13 (22.49) | -16.67 (19.25)
  Dyspnoea, Week 84: number analyzed (Participants) | 18 | 3
  Dyspnoea, Week 84 | -9.26 (25.06) | 0.00 (0.00)
  Dyspnoea, Week 93: number analyzed (Participants) | 20 | 2
  Dyspnoea, Week 93 | 0.00 (35.87) | -16.67 (23.57)
  Dyspnoea, Week 102: number analyzed (Participants) | 16 | 1
  Dyspnoea, Week 102 | 4.17 (26.87) | 0.00 (NA) — The standard deviation is a measure of the amount of variation or dispersion of a set of values. Number analyzed is 1 so standard deviation is not available.
  Dyspnoea, Week 111: number analyzed (Participants) | 13 | 0
  Dyspnoea, Week 111 | -7.69 (33.76) |
  Dyspnoea, Week 120: number analyzed (Participants) | 14 | 0
  Dyspnoea, Week 120 | 0.00 (22.65) |
  Dyspnoea, Week 129: number analyzed (Participants) | 14 | 0
  Dyspnoea, Week 129 | 2.38 (24.33) |
  Dyspnoea, Week 138: number analyzed (Participants) | 14 | 0
  Dyspnoea, Week 138 | -2.38 (27.62) |
  Dyspnoea, Week 147: number analyzed (Participants) | 14 | 0
  Dyspnoea, Week 147 | -4.76 (22.10) |
  Dyspnoea, Week 156: number analyzed (Participants) | 7 | 0
  Dyspnoea, Week 156 | 0.00 (19.25) |
  Dyspnoea, Week 165: number analyzed (Participants) | 8 | 0
  Dyspnoea, Week 165 | -4.17 (21.36) |
  Dyspnoea, Week 174: number analyzed (Participants) | 7 | 0
  Dyspnoea, Week 174 | 4.76 (23.00) |
  Dyspnoea, Week 183: number analyzed (Participants) | 5 | 0
  Dyspnoea, Week 183 | 6.67 (27.89) |
  Dyspnoea, Week 192: number analyzed (Participants) | 4 | 0
  Dyspnoea, Week 192 | 0.00 (27.22) |
  Dyspnoea, Week 201: number analyzed (Participants) | 1 | 0
  Dyspnoea, Week 201 | 0.00 (NA) — The standard deviation is a measure of the amount of variation or dispersion of a set of values. Number analyzed is 1 so standard deviation is not available. |
  Dyspnoea, Week 210: number analyzed (Participants) | 1 | 0
  Dyspnoea, Week 210 | 0.00 (NA) — The standard deviation is a measure of the amount of variation or dispersion of a set of values. Number analyzed is 1 so standard deviation is not available. |
  Dyspnoea, Safety Follow-Up Visit: number analyzed (Participants) | 11 | 12
  Dyspnoea, Safety Follow-Up Visit | 24.24 (44.95) | -2.78 (43.71)
  Insomnia, Baseline: number analyzed (Participants) | 294 | 146
  Insomnia, Baseline | 30.50 (29.97) | 31.05 (32.44)
  Insomnia, Week 6: number analyzed (Participants) | 222 | 115
  Insomnia, Week 6 | -1.95 (31.25) | -1.16 (33.60)
  Insomnia, Week 12: number analyzed (Participants) | 150 | 64
  Insomnia, Week 12 | -1.78 (31.32) | -3.65 (33.13)
  Insomnia, Week 18: number analyzed (Participants) | 122 | 40
  Insomnia, Week 18 | -4.37 (27.76) | -2.50 (36.51)
  Insomnia, Week 24: number analyzed (Participants) | 107 | 30
  Insomnia, Week 24 | -6.23 (29.01) | -5.56 (31.66)
  Insomnia, Week 30: number analyzed (Participants) | 84 | 23
  Insomnia, Week 30 | -3.17 (26.19) | -15.94 (28.19)
  Insomnia, Week 36: number analyzed (Participants) | 63 | 16
  Insomnia, Week 36 | -3.17 (26.58) | -18.75 (34.36)
  Insomnia, Week 42: number analyzed (Participants) | 54 | 14
  Insomnia, Week 42 | -3.09 (36.21) | -9.52 (27.51)
  Insomnia, Week 48: number analyzed (Participants) | 43 | 12
  Insomnia, Week 48 | -6.20 (27.46) | 2.78 (26.43)
  Insomnia, Week 57: number analyzed (Participants) | 37 | 8
  Insomnia, Week 57 | -9.91 (32.27) | 4.17 (33.03)
  Insomnia, Week 66: number analyzed (Participants) | 33 | 5
  Insomnia, Week 66 | -8.08 (27.68) | -6.67 (14.91)
  Insomnia, Week 75: number analyzed (Participants) | 26 | 4
  Insomnia, Week 75 | -8.97 (27.58) | -16.67 (19.25)
  Insomnia, Week 84: number analyzed (Participants) | 18 | 3
  Insomnia, Week 84 | -7.41 (24.40) | -22.22 (19.25)
  Insomnia, Week 93: number analyzed (Participants) | 20 | 2
  Insomnia, Week 93 | -8.33 (23.88) | 0.00 (0.00)
  Insomnia, Week 102: number analyzed (Participants) | 16 | 1
  Insomnia, Week 102 | -10.42 (20.07) | 0.00 (NA) — The standard deviation is a measure of the amount of variation or dispersion of a set of values. Number analyzed is 1 so standard deviation is not available.
  Insomnia, Week 111: number analyzed (Participants) | 14 | 0
  Insomnia, Week 111 | -9.52 (20.37) |
  Insomnia, Week 120: number analyzed (Participants) | 14 | 0
  Insomnia, Week 120 | -11.90 (21.11) |
  Insomnia, Week 129: number analyzed (Participants) | 14 | 0
  Insomnia, Week 129 | -9.52 (20.37) |
  Insomnia, Week 138: number analyzed (Participants) | 14 | 0
  Insomnia, Week 138 | -16.67 (21.68) |
  Insomnia, Week 147: number analyzed (Participants) | 14 | 0
  Insomnia, Week 147 | -14.29 (28.39) |
  Insomnia, Week 156: number analyzed (Participants) | 7 | 0
  Insomnia, Week 156 | -4.76 (12.60) |
  Insomnia, Week 165: number analyzed (Participants) | 8 | 0
  Insomnia, Week 165 | 0.00 (17.82) |
  Insomnia, Week 174: number analyzed (Participants) | 7 | 0
  Insomnia, Week 174 | -9.52 (16.27) |
  Insomnia, Week 183: number analyzed (Participants) | 5 | 0
  Insomnia, Week 183 | -13.33 (38.01) |
  Insomnia, Week 192: number analyzed (Participants) | 4 | 0
  Insomnia, Week 192 | -8.33 (16.67) |
  Insomnia, Week 201: number analyzed (Participants) | 2 | 0
  Insomnia, Week 201 | -33.33 (47.14) |
  Insomnia, Week 210: number analyzed (Participants) | 1 | 0
  Insomnia, Week 210 | -33.33 (NA) — The standard deviation is a measure of the amount of variation or dispersion of a set of values. Number analyzed is 1 so standard deviation is not available. |
  Insomnia, Safety Follow-Up Visit: number analyzed (Participants) | 11 | 13
  Insomnia, Safety Follow-Up Visit | 12.12 (42.88) | -5.13 (35.61)
  Appetite Loss, Baseline: number analyzed (Participants) | 294 | 146
  Appetite Loss, Baseline | 31.63 (33.06) | 31.05 (32.91)
  Appetite Loss, Week 6: number analyzed (Participants) | 221 | 114
  Appetite Loss, Week 6 | 1.06 (33.99) | 0.00 (38.40)
  Appetite Loss, Week 12: number analyzed (Participants) | 150 | 64
  Appetite Loss, Week 12 | -4.22 (35.46) | 7.29 (32.24)
  Appetite Loss, Week 18: number analyzed (Participants) | 122 | 40
  Appetite Loss, Week 18 | -7.38 (33.06) | 13.33 (27.01)
  Appetite Loss, Week 24: number analyzed (Participants) | 106 | 30
  Appetite Loss, Week 24 | -9.43 (28.27) | 10.00 (32.93)
  Appetite Loss, Week 30: number analyzed (Participants) | 84 | 23
  Appetite Loss, Week 30 | -12.30 (28.24) | 7.25 (31.71)
  Appetite Loss, Week 36: number analyzed (Participants) | 63 | 16
  Appetite Loss, Week 36 | -11.11 (33.87) | 6.25 (30.35)
  Appetite Loss, Week 42: number analyzed (Participants) | 54 | 14
  Appetite Loss, Week 42 | -7.41 (32.81) | 2.38 (27.62)
  Appetite Loss, Week 48: number analyzed (Participants) | 43 | 12
  Appetite Loss, Week 48 | -10.85 (29.74) | 5.56 (44.57)
  Appetite Loss, Week 57: number analyzed (Participants) | 37 | 8
  Appetite Loss, Week 57 | -6.31 (31.27) | 8.33 (42.72)
  Appetite Loss, Week 66: number analyzed (Participants) | 33 | 5
  Appetite Loss, Week 66 | -9.09 (29.19) | 13.33 (29.81)
  Appetite Loss, Week 75: number analyzed (Participants) | 26 | 4
  Appetite Loss, Week 75 | -10.26 (30.94) | 0.00 (27.22)
  Appetite Loss, Week 84: number analyzed (Participants) | 19 | 3
  Appetite Loss, Week 84 | -17.54 (28.04) | 22.22 (19.25)
  Appetite Loss, Week 93: number analyzed (Participants) | 20 | 2
  Appetite Loss, Week 93 | -10.00 (26.71) | 50.00 (23.57)
  Appetite Loss, Week 102: number analyzed (Participants) | 16 | 1
  Appetite Loss, Week 102 | -10.42 (20.07) | 66.67 (NA) — The standard deviation is a measure of the amount of variation or dispersion of a set of values. Number analyzed is 1 so standard deviation is not available.
  Appetite Loss, Week 111: number analyzed (Participants) | 14 | 0
  Appetite Loss, Week 111 | -7.14 (23.31) |
  Appetite Loss, Week 120: number analyzed (Participants) | 14 | 0
  Appetite Loss, Week 120 | -9.52 (27.51) |
  Appetite Loss, Week 129: number analyzed (Participants) | 14 | 0
  Appetite Loss, Week 129 | -7.14 (23.31) |
  Appetite Loss, Week 138: number analyzed (Participants) | 14 | 0
  Appetite Loss, Week 138 | -9.52 (24.21) |
  Appetite Loss, Week 147: number analyzed (Participants) | 14 | 0
  Appetite Loss, Week 147 | -16.67 (31.35) |
  Appetite Loss, Week 156: number analyzed (Participants) | 7 | 0
  Appetite Loss, Week 156 | 0.00 (0.00) |
  Appetite Loss, Week 165: number analyzed (Participants) | 8 | 0
  Appetite Loss, Week 165 | 0.00 (0.00) |
  Appetite Loss, Week 174: number analyzed (Participants) | 7 | 0
  Appetite Loss, Week 174 | -9.52 (25.20) |
  Appetite Loss, Week 183: number analyzed (Participants) | 5 | 0
  Appetite Loss, Week 183 | -13.33 (29.81) |
  Appetite Loss, Week 192: number analyzed (Participants) | 4 | 0
  Appetite Loss, Week 192 | 8.33 (16.67) |
  Appetite Loss, Week 201: number analyzed (Participants) | 2 | 0
  Appetite Loss, Week 201 | 16.67 (23.57) |
  Appetite Loss, Week 210: number analyzed (Participants) | 1 | 0
  Appetite Loss, Week 210 | 0.00 (NA) — The standard deviation is a measure of the amount of variation or dispersion of a set of values. Number analyzed is 1 so standard deviation is not available. |
  Appetite Loss, Safety Follow-Up Visit: number analyzed (Participants) | 11 | 13
  Appetite Loss, Safety Follow-Up Visit | -9.09 (39.70) | -7.69 (52.97)
  Constipation, Baseline: number analyzed (Participants) | 294 | 146
  Constipation, Baseline | 21.20 (30.67) | 21.92 (27.80)
  Constipation, Week 6: number analyzed (Participants) | 221 | 115
  Constipation, Week 6 | -0.45 (27.98) | 1.45 (31.65)
  Constipation, Week 12: number analyzed (Participants) | 149 | 64
  Constipation, Week 12 | -2.46 (29.79) | -0.52 (28.17)
  Constipation, Week 18: number analyzed (Participants) | 122 | 40
  Constipation, Week 18 | -6.01 (29.39) | 0.83 (29.71)
  Constipation, Week 24: number analyzed (Participants) | 107 | 30
  Constipation, Week 24 | -5.61 (29.13) | 1.11 (22.29)
  Constipation, Week 30: number analyzed (Participants) | 84 | 23
  Constipation, Week 30 | -6.75 (27.76) | 5.80 (25.92)
  Constipation, Week 36: number analyzed (Participants) | 63 | 16
  Constipation, Week 36 | -7.94 (33.18) | 6.25 (18.13)
  Constipation, Week 42: number analyzed (Participants) | 54 | 14
  Constipation, Week 42 | -4.94 (31.33) | 0.00 (18.49)
  Constipation, Week 48: number analyzed (Participants) | 44 | 11
  Constipation, Week 48 | -10.61 (32.76) | -6.06 (25.03)
  Constipation, Week 57: number analyzed (Participants) | 37 | 8
  Constipation, Week 57 | -15.32 (28.97) | -8.33 (15.43)
  Constipation, Week 66: number analyzed (Participants) | 33 | 5
  Constipation, Week 66 | -13.13 (27.56) | 0.00 (23.57)
  Constipation, Week 75: number analyzed (Participants) | 26 | 4
  Constipation, Week 75 | -5.13 (32.24) | 16.67 (57.74)
  Constipation, Week 84: number analyzed (Participants) | 19 | 3
  Constipation, Week 84 | -3.51 (31.22) | 11.11 (38.49)
  Constipation, Week 93: number analyzed (Participants) | 20 | 2
  Constipation, Week 93 | -8.33 (35.66) | 33.33 (0.00)
  Constipation, Week 102: number analyzed (Participants) | 16 | 1
  Constipation, Week 102 | -10.42 (35.94) | 33.33 (NA) — The standard deviation is a measure of the amount of variation or dispersion of a set of values. Number analyzed is 1 so standard deviation is not available.
  Constipation, Week 111: number analyzed (Participants) | 14 | 0
  Constipation, Week 111 | -7.14 (41.71) |
  Constipation, Week 120: number analyzed (Participants) | 14 | 0
  Constipation, Week 120 | -4.76 (41.05) |
  Constipation, Week 129: number analyzed (Participants) | 14 | 0
  Constipation, Week 129 | -7.14 (41.71) |
  Constipation, Week 138: number analyzed (Participants) | 14 | 0
  Constipation, Week 138 | -9.52 (47.91) |
  Constipation, Week 147: number analyzed (Participants) | 14 | 0
  Constipation, Week 147 | -11.90 (42.58) |
  Constipation, Week 156: number analyzed (Participants) | 7 | 0
  Constipation, Week 156 | -14.29 (26.23) |
  Constipation, Week 165: number analyzed (Participants) | 8 | 0
  Constipation, Week 165 | -8.33 (29.55) |
  Constipation, Week 174: number analyzed (Participants) | 7 | 0
  Constipation, Week 174 | -14.29 (26.23) |
  Constipation, Week 183: number analyzed (Participants) | 5 | 0
  Constipation, Week 183 | -13.33 (18.26) |
  Constipation, Week 192: number analyzed (Participants) | 4 | 0
  Constipation, Week 192 | 0.00 (27.22) |
  Constipation, Week 201: number analyzed (Participants) | 2 | 0
  Constipation, Week 201 | 16.67 (23.57) |
  Constipation, Week 210: number analyzed (Participants) | 1 | 0
  Constipation, Week 210 | 0.00 (NA) — The standard deviation is a measure of the amount of variation or dispersion of a set of values. Number analyzed is 1 so standard deviation is not available. |
  Constipation, Safety Follow-Up Visit: number analyzed (Participants) | 11 | 13
  Constipation, Safety Follow-Up Visit | 3.03 (45.84) | 7.69 (30.89)
  Diarrhoea, Baseline: number analyzed (Participants) | 290 | 146
  Diarrhoea, Baseline | 5.63 (15.28) | 5.71 (16.31)
  Diarrhoea, Week 6: number analyzed (Participants) | 219 | 115
  Diarrhoea, Week 6 | -0.61 (19.93) | 3.48 (23.93)
  Diarrhoea, Week 12: number analyzed (Participants) | 148 | 63
  Diarrhoea, Week 12 | 1.80 (21.57) | 1.06 (18.90)
  Diarrhoea, Week 18: number analyzed (Participants) | 120 | 40
  Diarrhoea, Week 18 | -0.83 (18.57) | 5.83 (24.91)
  Diarrhoea, Week 24: number analyzed (Participants) | 104 | 30
  Diarrhoea, Week 24 | 0.00 (18.58) | 5.56 (17.69)
  Diarrhoea, Week 30: number analyzed (Participants) | 83 | 23
  Diarrhoea, Week 30 | 2.01 (19.02) | 4.35 (11.48)
  Diarrhoea, Week 36: number analyzed (Participants) | 62 | 16
  Diarrhoea, Week 36 | 0.00 (20.91) | 2.08 (8.33)
  Diarrhoea, Week 42: number analyzed (Participants) | 54 | 14
  Diarrhoea, Week 42 | -3.09 (17.46) | 2.38 (8.91)
  Diarrhoea, Week 48: number analyzed (Participants) | 44 | 12
  Diarrhoea, Week 48 | -0.76 (15.23) | 8.33 (20.72)
  Diarrhoea, Week 57: number analyzed (Participants) | 37 | 8
  Diarrhoea, Week 57 | 0.00 (20.79) | 4.17 (11.79)
  Diarrhoea, Week 66: number analyzed (Participants) | 33 | 5
  Diarrhoea, Week 66 | -4.04 (18.18) | 6.67 (14.91)
  Diarrhoea, Week 75: number analyzed (Participants) | 26 | 4
  Diarrhoea, Week 75 | -5.13 (15.47) | 0.00 (0.00)
  Diarrhoea, Week 84: number analyzed (Participants) | 19 | 3
  Diarrhoea, Week 84 | 1.75 (13.49) | 0.00 (0.00)
  Diarrhoea, Week 93: number analyzed (Participants) | 20 | 2
  Diarrhoea, Week 93 | 1.67 (25.31) | 0.00 (0.00)
  Diarrhoea, Week 102: number analyzed (Participants) | 16 | 1
  Diarrhoea, Week 102 | 0.00 (17.21) | 0.00 (NA) — The standard deviation is a measure of the amount of variation or dispersion of a set of values. Number analyzed is 1 so standard deviation is not available.
  Diarrhoea, Week 111: number analyzed (Participants) | 14 | 0
  Diarrhoea, Week 111 | 7.14 (29.75) |
  Diarrhoea, Week 120: number analyzed (Participants) | 14 | 0
  Diarrhoea, Week 120 | 4.76 (34.24) |
  Diarrhoea, Week 129: number analyzed (Participants) | 14 | 0
  Diarrhoea, Week 129 | 2.38 (33.24) |
  Diarrhoea, Week 138: number analyzed (Participants) | 14 | 0
  Diarrhoea, Week 138 | -4.76 (17.82) |
  Diarrhoea, Week 147: number analyzed (Participants) | 14 | 0
  Diarrhoea, Week 147 | -4.76 (22.10) |
  Diarrhoea, Week 156: number analyzed (Participants) | 7 | 0
  Diarrhoea, Week 156 | -4.76 (12.60) |
  Diarrhoea, Week 165: number analyzed (Participants) | 7 | 0
  Diarrhoea, Week 165 | 0.00 (0.00) |
  Diarrhoea, Week 174: number analyzed (Participants) | 7 | 0
  Diarrhoea, Week 174 | -9.52 (25.20) |
  Diarrhoea, Week 183: number analyzed (Participants) | 5 | 0
  Diarrhoea, Week 183 | -13.33 (29.81) |
  Diarrhoea, Week 192: number analyzed (Participants) | 4 | 0
  Diarrhoea, Week 192 | 0.00 (0.00) |
  Diarrhoea, Week 201: number analyzed (Participants) | 2 | 0
  Diarrhoea, Week 201 | 0.00 (0.00) |
  Diarrhoea, Week 210: number analyzed (Participants) | 1 | 0
  Diarrhoea, Week 210 | 0.00 (NA) — The standard deviation is a measure of the amount of variation or dispersion of a set of values. Number analyzed is 1 so standard deviation is not available. |
  Diarrhoea, Safety Follow-Up Visit: number analyzed (Participants) | 11 | 13
  Diarrhoea, Safety Follow-Up Visit | 6.06 (29.13) | 0.00 (13.61)
  Financial Difficulties, Baseline: number analyzed (Participants) | 291 | 146
  Financial Difficulties, Baseline | 22.22 (28.81) | 20.32 (28.60)
  Financial Difficulties, Week 6: number analyzed (Participants) | 219 | 115
  Financial Difficulties, Week 6 | -3.20 (27.00) | 0.00 (25.74)
  Financial Difficulties, Week 12: number analyzed (Participants) | 148 | 64
  Financial Difficulties, Week 12 | -4.95 (27.59) | 1.56 (26.18)
  Financial Difficulties, Week 18: number analyzed (Participants) | 121 | 40
  Financial Difficulties, Week 18 | -4.41 (23.94) | 4.17 (27.41)
  Financial Difficulties, Week 24: number analyzed (Participants) | 105 | 30
  Financial Difficulties, Week 24 | -4.76 (30.11) | 2.22 (23.05)
  Financial Difficulties, Week 30: number analyzed (Participants) | 83 | 23
  Financial Difficulties, Week 30 | -3.21 (24.20) | -1.45 (23.52)
  Financial Difficulties, Week 36: number analyzed (Participants) | 62 | 15
  Financial Difficulties, Week 36 | -2.69 (28.50) | 4.44 (21.33)
  Financial Difficulties, Week 42: number analyzed (Participants) | 54 | 14
  Financial Difficulties, Week 42 | -1.85 (33.28) | 2.38 (27.62)
  Financial Difficulties, Week 48: number analyzed (Participants) | 44 | 12
  Financial Difficulties, Week 48 | -0.76 (29.19) | -5.56 (27.83)
  Financial Difficulties, Week 57: number analyzed (Participants) | 37 | 8
  Financial Difficulties, Week 57 | -4.50 (32.55) | -4.17 (21.36)
  Financial Difficulties, Week 66: number analyzed (Participants) | 33 | 5
  Financial Difficulties, Week 66 | 0.00 (28.87) | -6.67 (27.89)
  Financial Difficulties, Week 75: number analyzed (Participants) | 26 | 4
  Financial Difficulties, Week 75 | 1.28 (29.03) | 8.33 (31.91)
  Financial Difficulties, Week 84: number analyzed (Participants) | 19 | 3
  Financial Difficulties, Week 84 | 3.51 (26.98) | -22.22 (19.25)
  Financial Difficulties, Week 93: number analyzed (Participants) | 20 | 2
  Financial Difficulties, Week 93 | 0.00 (26.49) | -16.67 (23.57)
  Financial Difficulties, Week 102: number analyzed (Participants) | 16 | 1
  Financial Difficulties, Week 102 | 2.08 (25.73) | -33.33 (NA) — The standard deviation is a measure of the amount of variation or dispersion of a set of values. Number analyzed is 1 so standard deviation is not available.
  Financial Difficulties, Week 111: number analyzed (Participants) | 14 | 0
  Financial Difficulties, Week 111 | 2.38 (27.62) |
  Financial Difficulties, Week 120: number analyzed (Participants) | 14 | 0
  Financial Difficulties, Week 120 | -2.38 (27.62) |
  Financial Difficulties, Week 129: number analyzed (Participants) | 14 | 0
  Financial Difficulties, Week 129 | -2.38 (24.33) |
  Financial Difficulties, Week 138: number analyzed (Participants) | 14 | 0
  Financial Difficulties, Week 138 | 2.38 (30.56) |
  Financial Difficulties, Week 147: number analyzed (Participants) | 14 | 0
  Financial Difficulties, Week 147 | -2.38 (27.62) |
  Financial Difficulties, Week 156: number analyzed (Participants) | 7 | 0
  Financial Difficulties, Week 156 | -9.52 (31.71) |
  Financial Difficulties, Week 165: number analyzed (Participants) | 8 | 0
  Financial Difficulties, Week 165 | 4.17 (37.53) |
  Financial Difficulties, Week 174: number analyzed (Participants) | 7 | 0
  Financial Difficulties, Week 174 | -9.52 (31.71) |
  Financial Difficulties, Week 183: number analyzed (Participants) | 5 | 0
  Financial Difficulties, Week 183 | 0.00 (23.57) |
  Financial Difficulties, Week 192: number analyzed (Participants) | 4 | 0
  Financial Difficulties, Week 192 | 0.00 (27.22) |
  Financial Difficulties, Week 201: number analyzed (Participants) | 2 | 0
  Financial Difficulties, Week 201 | 16.67 (23.57) |
  Financial Difficulties, Week 210: number analyzed (Participants) | 1 | 0
  Financial Difficulties, Week 210 | 0.00 (NA) — The standard deviation is a measure of the amount of variation or dispersion of a set of values. Number analyzed is 1 so standard deviation is not available. |
  Financial Difficulties, Safety Follow-Up Visit: number analyzed (Participants) | 11 | 13
  Financial Difficulties, Safety Follow-Up Visit | -3.03 (43.34) | 0.00 (27.22)

8. Secondary Outcome: Change From Baseline in EORTC QLQ Supplementary Lung Cancer Module 13 (EORTC QLQ-LC13) Score
Description: The EORTC QLQ-LC13 module incorporates one multiple item scale to assess dyspnea and a series of single items assessing pain, coughing, sore mouth, dysphagia, peripheral neuropathy, alopecia, and hemoptysis. The EORTC QLQ-LC13 was scored according to the EORTC scoring manual (Fayers et al. 2001). All EORTC scales and single-item measures are linearly transformed so that each score has a range of 0-100. A high score for a functional/global health status scale represents a high or healthy level of functioning/HRQoL (Health-Related Quality of Life); however, a high score for a symptom scale or item represents a high level of symptomatology or problems. A≥10-point change in the symptoms subscale score was perceived by participants as clinically significant (Osoba et al. 1998). A positive change from baseline indicates improvement and negative change from baseline indicated worsening.
Time Frame: as for outcome 7
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: units of a scale
Arm/Group | Atezolizumab | Single Agent Chemotherapy (Vinorelbine or Gemcitabine)
Number analyzed (Participants) | 302 | 151
units of a scale
  Dyspnoea, Baseline: number analyzed (Participants) | 287 | 140
  Dyspnoea, Baseline | 34.30 (25.69) | 36.67 (25.35)
  Dyspnoea, Week 6: number analyzed (Participants) | 207 | 109
  Dyspnoea, Week 6 | 1.13 (19.90) | 0.92 (24.25)
  Dyspnoea, Week 12: number analyzed (Participants) | 144 | 62
  Dyspnoea, Week 12 | -0.23 (24.28) | -2.87 (24.55)
  Dyspnoea, Week 18: number analyzed (Participants) | 114 | 37
  Dyspnoea, Week 18 | -4.78 (18.93) | 0.90 (23.33)
  Dyspnoea, Week 24: number analyzed (Participants) | 99 | 29
  Dyspnoea, Week 24 | -5.05 (22.91) | 2.68 (23.13)
  Dyspnoea, Week 30: number analyzed (Participants) | 79 | 22
  Dyspnoea, Week 30 | -5.34 (22.00) | 1.52 (25.03)
  Dyspnoea, Week 36: number analyzed (Participants) | 57 | 14
  Dyspnoea, Week 36 | -3.90 (26.85) | 5.56 (19.85)
  Dyspnoea, Week 42: number analyzed (Participants) | 48 | 13
  Dyspnoea, Week 42 | -11.11 (26.63) | -6.84 (22.01)
  Dyspnoea, Week 48: number analyzed (Participants) | 39 | 12
  Dyspnoea, Week 48 | -4.84 (26.83) | 1.85 (22.64)
  Dyspnoea, Week 57: number analyzed (Participants) | 31 | 8
  Dyspnoea, Week 57 | -7.89 (20.53) | 4.17 (15.64)
  Dyspnoea, Week 66: number analyzed (Participants) | 27 | 5
  Dyspnoea, Week 66 | -6.58 (24.12) | 0.00 (13.61)
  Dyspnoea, Week 75: number analyzed (Participants) | 22 | 4
  Dyspnoea, Week 75 | -4.55 (23.67) | -2.78 (30.60)
  Dyspnoea, Week 84: number analyzed (Participants) | 17 | 3
  Dyspnoea, Week 84 | -8.50 (23.74) | 3.70 (23.13)
  Dyspnoea, Week 93: number analyzed (Participants) | 19 | 2
  Dyspnoea, Week 93 | -2.34 (27.61) | 5.56 (7.86)
  Dyspnoea, Week 102: number analyzed (Participants) | 15 | 1
  Dyspnoea, Week 102 | -2.96 (21.19) | 0.00 (NA) — The standard deviation is a measure of the amount of variation or dispersion of a set of values. Number analyzed is 1 so standard deviation is not available.
  Dyspnoea, Week 111: number analyzed (Participants) | 13 | 0
  Dyspnoea, Week 111 | -2.56 (26.51) |
  Dyspnoea, Week 120: number analyzed (Participants) | 13 | 0
  Dyspnoea, Week 120 | -4.27 (24.23) |
  Dyspnoea, Week 129: number analyzed (Participants) | 12 | 0
  Dyspnoea, Week 129 | 3.70 (15.95) |
  Dyspnoea, Week 138: number analyzed (Participants) | 13 | 0
  Dyspnoea, Week 138 | 0.00 (24.43) |
  Dyspnoea, Week 147: number analyzed (Participants) | 13 | 0
  Dyspnoea, Week 147 | -0.85 (26.24) |
  Dyspnoea, Week 156: number analyzed (Participants) | 7 | 0
  Dyspnoea, Week 156 | 1.59 (14.95) |
  Dyspnoea, Week 165: number analyzed (Participants) | 6 | 0
  Dyspnoea, Week 165 | -1.85 (21.56) |
  Dyspnoea, Week 174: number analyzed (Participants) | 7 | 0
  Dyspnoea, Week 174 | 1.59 (17.48) |
  Dyspnoea, Week 183: number analyzed (Participants) | 4 | 0
  Dyspnoea, Week 183 | 5.56 (21.28) |
  Dyspnoea, Week 192: number analyzed (Participants) | 4 | 0
  Dyspnoea, Week 192 | 5.56 (26.45) |
  Dyspnoea, Week 201: number analyzed (Participants) | 2 | 0
  Dyspnoea, Week 201 | 0.00 (15.71) |
  Dyspnoea, Week 210: number analyzed (Participants) | 1 | 0
  Dyspnoea, Week 210 | 0.00 (NA) — The standard deviation is a measure of the amount of variation or dispersion of a set of values. Number analyzed is 1 so standard deviation is not available. |
  Dyspnoea, Safety Follow-Up Visit: number analyzed (Participants) | 11 | 12
  Dyspnoea, Safety Follow-Up Visit | 12.12 (29.17) | 6.48 (31.94)
  Coughing, Baseline: number analyzed (Participants) | 295 | 147
  Coughing, Baseline | 41.36 (30.24) | 46.26 (28.25)
  Coughing, Week 6: number analyzed (Participants) | 222 | 116
  Coughing, Week 6 | -1.80 (25.10) | -5.46 (29.80)
  Coughing, Week 12: number analyzed (Participants) | 149 | 64
  Coughing, Week 12 | -7.61 (30.79) | -9.38 (29.97)
  Coughing, Week 18: number analyzed (Participants) | 121 | 39
  Coughing, Week 18 | -9.64 (29.01) | -3.42 (34.87)
  Coughing, Week 24: number analyzed (Participants) | 106 | 30
  Coughing, Week 24 | -11.01 (30.42) | 3.33 (30.76)
  Coughing, Week 30: number analyzed (Participants) | 83 | 24
  Coughing, Week 30 | -9.24 (33.46) | 0.00 (26.01)
  Coughing, Week 36: number analyzed (Participants) | 61 | 16
  Coughing, Week 36 | -7.10 (35.02) | 0.00 (34.43)
  Coughing, Week 42: number analyzed (Participants) | 53 | 14
  Coughing, Week 42 | -10.06 (31.07) | -2.38 (27.62)
  Coughing, Week 48: number analyzed (Participants) | 44 | 12
  Coughing, Week 48 | -15.91 (30.06) | 0.00 (20.10)
  Coughing, Week 57: number analyzed (Participants) | 35 | 8
  Coughing, Week 57 | -14.29 (31.61) | 4.17 (27.82)
  Coughing, Week 66: number analyzed (Participants) | 32 | 5
  Coughing, Week 66 | -11.46 (33.45) | -13.33 (18.26)
  Coughing, Week 75: number analyzed (Participants) | 25 | 4
  Coughing, Week 75 | -9.33 (28.09) | -8.33 (16.67)
  Coughing, Week 84: number analyzed (Participants) | 19 | 3
  Coughing, Week 84 | -19.30 (32.04) | 11.11 (19.25)
  Coughing, Week 93: number analyzed (Participants) | 20 | 2
  Coughing, Week 93 | -21.67 (31.11) | 16.67 (23.57)
  Coughing, Week 102: number analyzed (Participants) | 16 | 1
  Coughing, Week 102 | -14.58 (20.97) | 0.00 (NA) — The standard deviation is a measure of the amount of variation or dispersion of a set of values. Number analyzed is 1 so standard deviation is not available.
  Coughing, Week 111: number analyzed (Participants) | 14 | 0
  Coughing, Week 111 | -11.90 (21.11) |
  Coughing, Week 120: number analyzed (Participants) | 14 | 0
  Coughing, Week 120 | -11.90 (21.11) |
  Coughing, Week 129: number analyzed (Participants) | 14 | 0
  Coughing, Week 129 | -14.29 (21.54) |
  Coughing, Week 138: number analyzed (Participants) | 14 | 0
  Coughing, Week 138 | -16.67 (21.68) |
  Coughing, Week 147: number analyzed (Participants) | 14 | 0
  Coughing, Week 147 | -21.43 (24.83) |
  Coughing, Week 156: number analyzed (Participants) | 7 | 0
  Coughing, Week 156 | -23.81 (31.71) |
  Coughing, Week 165: number analyzed (Participants) | 8 | 0
  Coughing, Week 165 | -16.67 (35.63) |
  Coughing, Week 174: number analyzed (Participants) | 7 | 0
  Coughing, Week 174 | -19.05 (32.53) |
  Coughing, Week 183: number analyzed (Participants) | 4 | 0
  Coughing, Week 183 | 0.00 (27.22) |
  Coughing, Week 192: number analyzed (Participants) | 4 | 0
  Coughing, Week 192 | -16.67 (19.25) |
  Coughing, Week 201: number analyzed (Participants) | 2 | 0
  Coughing, Week 201 | 0.00 (0.00) |
  Coughing, Week 210: number analyzed (Participants) | 1 | 0
  Coughing, Week 210 | 0.00 (NA) — The standard deviation is a measure of the amount of variation or dispersion of a set of values. Number analyzed is 1 so standard deviation is not available. |
  Coughing, Safety Follow-Up Visit: number analyzed (Participants) | 11 | 13
  Coughing, Safety Follow-Up Visit | 3.03 (37.87) | -17.95 (25.88)
  Haemoptysis, Baseline: number analyzed (Participants) | 296 | 146
  Haemoptysis, Baseline | 5.86 (14.38) | 7.76 (18.79)
  Haemoptysis, Week 6: number analyzed (Participants) | 223 | 115
  Haemoptysis, Week 6 | 0.75 (19.10) | -4.64 (21.58)
  Haemoptysis, Week 12: number analyzed (Participants) | 148 | 63
  Haemoptysis, Week 12 | -1.80 (15.45) | -3.17 (20.49)
  Haemoptysis, Week 18: number analyzed (Participants) | 122 | 39
  Haemoptysis, Week 18 | -1.64 (15.95) | -1.71 (17.01)
  Haemoptysis, Week 24: number analyzed (Participants) | 106 | 30
  Haemoptysis, Week 24 | -2.52 (13.57) | -1.11 (18.54)
  Haemoptysis, Week 30: number analyzed (Participants) | 84 | 23
  Haemoptysis, Week 30 | -3.97 (14.08) | -2.90 (13.90)
  Haemoptysis, Week 36: number analyzed (Participants) | 60 | 16
  Haemoptysis, Week 36 | -1.67 (17.81) | -6.25 (18.13)
  Haemoptysis, Week 42: number analyzed (Participants) | 53 | 14
  Haemoptysis, Week 42 | -1.26 (15.96) | -2.38 (20.52)
  Haemoptysis, Week 48: number analyzed (Participants) | 44 | 12
  Haemoptysis, Week 48 | -3.79 (12.89) | -5.56 (19.25)
  Haemoptysis, Week 57: number analyzed (Participants) | 36 | 8
  Haemoptysis, Week 57 | -2.78 (18.47) | -8.33 (23.57)
  Haemoptysis, Week 66: number analyzed (Participants) | 31 | 5
  Haemoptysis, Week 66 | -2.15 (11.97) | 0.00 (0.00)
  Haemoptysis, Week 75: number analyzed (Participants) | 25 | 4
  Haemoptysis, Week 75 | -1.33 (11.71) | 0.00 (0.00)
  Haemoptysis, Week 84: number analyzed (Participants) | 19 | 3
  Haemoptysis, Week 84 | -3.51 (10.51) | 0.00 (0.00)
  Haemoptysis, Week 93: number analyzed (Participants) | 20 | 2
  Haemoptysis, Week 93 | -1.67 (13.13) | 0.00 (0.00)
  Haemoptysis, Week 102: number analyzed (Participants) | 16 | 1
  Haemoptysis, Week 102 | -2.08 (8.33) | 0.00 (NA) — The standard deviation is a measure of the amount of variation or dispersion of a set of values. Number analyzed is 1 so standard deviation is not available.
  Haemoptysis, Week 111: number analyzed (Participants) | 14 | 0
  Haemoptysis, Week 111 | -2.38 (8.91) |
  Haemoptysis, Week 120: number analyzed (Participants) | 14 | 0
  Haemoptysis, Week 120 | -2.38 (8.91) |
  Haemoptysis, Week 129: number analyzed (Participants) | 14 | 0
  Haemoptysis, Week 129 | -2.38 (8.91) |
  Haemoptysis, Week 138: number analyzed (Participants) | 14 | 0
  Haemoptysis, Week 138 | -2.38 (8.91) |
  Haemoptysis, Week 147: number analyzed (Participants) | 14 | 0
  Haemoptysis, Week 147 | -2.38 (8.91) |
  Haemoptysis, Week 156: number analyzed (Participants) | 7 | 0
  Haemoptysis, Week 156 | 0.00 (0.00) |
  Haemoptysis, Week 165: number analyzed (Participants) | 8 | 0
  Haemoptysis, Week 165 | 0.00 (0.00) |
  Haemoptysis, Week 174: number analyzed (Participants) | 7 | 0
  Haemoptysis, Week 174 | 0.00 (0.00) |
  Haemoptysis, Week 183: number analyzed (Participants) | 4 | 0
  Haemoptysis, Week 183 | 0.00 (0.00) |
  Haemoptysis, Week 192: number analyzed (Participants) | 4 | 0
  Haemoptysis, Week 192 | 0.00 (0.00) |
  Haemoptysis, Week 201: number analyzed (Participants) | 2 | 0
  Haemoptysis, Week 201 | 0.00 (0.00) |
  Haemoptysis, Week 210: number analyzed (Participants) | 1 | 0
  Haemoptysis, Week 210 | 0.00 (NA) — The standard deviation is a measure of the amount of variation or dispersion of a set of values. Number analyzed is 1 so standard deviation is not available. |
  Haemoptysis, Safety Follow-Up Visit: number analyzed (Participants) | 11 | 13
  Haemoptysis, Safety Follow-Up Visit | 3.03 (17.98) | -2.56 (16.45)
  Sore Mouth, Baseline: number analyzed (Participants) | 296 | 146
  Sore Mouth, Baseline | 4.17 (13.50) | 5.02 (14.83)
  Sore Mouth, Week 6: number analyzed (Participants) | 223 | 115
  Sore Mouth, Week 6 | 1.64 (19.30) | 0.00 (20.23)
  Sore Mouth, Week 12: number analyzed (Participants) | 150 | 64
  Sore Mouth, Week 12 | -0.22 (17.91) | 0.00 (16.80)
  Sore Mouth, Week 18: number analyzed (Participants) | 122 | 39
  Sore Mouth, Week 18 | -0.82 (16.85) | 2.56 (20.78)
  Sore Mouth, Week 24: number analyzed (Participants) | 105 | 29
  Sore Mouth, Week 24 | -1.90 (19.52) | 2.30 (17.66)
  Sore Mouth, Week 30: number analyzed (Participants) | 84 | 23
  Sore Mouth, Week 30 | -3.57 (21.96) | 0.00 (17.41)
  Sore Mouth, Week 36: number analyzed (Participants) | 61 | 16
  Sore Mouth, Week 36 | -2.73 (22.19) | -2.08 (19.12)
  Sore Mouth, Week 42: number analyzed (Participants) | 53 | 14
  Sore Mouth, Week 42 | 0.00 (29.24) | 4.76 (28.81)
  Sore Mouth, Week 48: number analyzed (Participants) | 44 | 12
  Sore Mouth, Week 48 | -5.30 (18.94) | -2.78 (22.29)
  Sore Mouth, Week 57: number analyzed (Participants) | 36 | 8
  Sore Mouth, Week 57 | -5.56 (20.31) | 0.00 (17.82)
  Sore Mouth, Week 66: number analyzed (Participants) | 32 | 5
  Sore Mouth, Week 66 | -4.17 (16.40) | 6.67 (14.91)
  Sore Mouth, Week 75: number analyzed (Participants) | 25 | 4
  Sore Mouth, Week 75 | -5.33 (15.75) | 16.67 (19.25)
  Sore Mouth, Week 84: number analyzed (Participants) | 19 | 3
  Sore Mouth, Week 84 | -1.75 (7.65) | 11.11 (19.25)
  Sore Mouth, Week 93: number analyzed (Participants) | 20 | 2
  Sore Mouth, Week 93 | -1.67 (7.45) | 0.00 (0.00)
  Sore Mouth, Week 102: number analyzed (Participants) | 16 | 1
  Sore Mouth, Week 102 | 2.08 (8.33) | 0.00 (NA) — The standard deviation is a measure of the amount of variation or dispersion of a set of values. Number analyzed is 1 so standard deviation is not available.
  Sore Mouth, Week 111: number analyzed (Participants) | 14 | 0
  Sore Mouth, Week 111 | 0.00 (22.65) |
  Sore Mouth, Week 120: number analyzed (Participants) | 14 | 0
  Sore Mouth, Week 120 | 2.38 (8.91) |
  Sore Mouth, Week 129: number analyzed (Participants) | 14 | 0
  Sore Mouth, Week 129 | -4.76 (17.82) |
  Sore Mouth, Week 138: number analyzed (Participants) | 14 | 0
  Sore Mouth, Week 138 | 2.38 (8.91) |
  Sore Mouth, Week 147: number analyzed (Participants) | 14 | 0
  Sore Mouth, Week 147 | 0.00 (0.00) |
  Sore Mouth, Week 156: number analyzed (Participants) | 7 | 0
  Sore Mouth, Week 156 | 0.00 (0.00) |
  Sore Mouth, Week 165: number analyzed (Participants) | 8 | 0
  Sore Mouth, Week 165 | 4.17 (27.82) |
  Sore Mouth, Week 174: number analyzed (Participants) | 7 | 0
  Sore Mouth, Week 174 | 0.00 (0.00) |
  Sore Mouth, Week 183: number analyzed (Participants) | 4 | 0
  Sore Mouth, Week 183 | 0.00 (0.00) |
  Sore Mouth, Week 192: number analyzed (Participants) | 4 | 0
  Sore Mouth, Week 192 | 0.00 (0.00) |
  Sore Mouth, Week 201: number analyzed (Participants) | 2 | 0
  Sore Mouth, Week 201 | 0.00 (0.00) |
  Sore Mouth, Week 210: number analyzed (Participants) | 1 | 0
  Sore Mouth, Week 210 | 0.00 (NA) — The standard deviation is a measure of the amount of variation or dispersion of a set of values. Number analyzed is 1 so standard deviation is not available. |
  Sore Mouth, Safety Follow-Up Visit: number analyzed (Participants) | 11 | 13
  Sore Mouth, Safety Follow-Up Visit | 27.27 (32.72) | 0.00 (19.25)
  Dysphagia, Baseline: number analyzed (Participants) | 296 | 146
  Dysphagia, Baseline | 11.15 (23.60) | 8.68 (19.60)
  Dysphagia, Week 6: number analyzed (Participants) | 223 | 115
  Dysphagia, Week 6 | -1.20 (20.47) | 2.90 (25.96)
  Dysphagia, Week 12: number analyzed (Participants) | 151 | 64
  Dysphagia, Week 12 | -0.44 (21.77) | -1.04 (23.73)
  Dysphagia, Week 18: number analyzed (Participants) | 122 | 39
  Dysphagia, Week 18 | -2.19 (23.37) | -0.85 (29.11)
  Dysphagia, Week 24: number analyzed (Participants) | 106 | 30
  Dysphagia, Week 24 | -4.72 (23.20) | 1.11 (28.34)
  Dysphagia, Week 30: number analyzed (Participants) | 84 | 23
  Dysphagia, Week 30 | -3.57 (23.15) | 2.90 (28.27)
  Dysphagia, Week 36: number analyzed (Participants) | 60 | 16
  Dysphagia, Week 36 | -6.11 (28.45) | 6.25 (13.44)
  Dysphagia, Week 42: number analyzed (Participants) | 53 | 14
  Dysphagia, Week 42 | -7.55 (31.11) | 4.76 (17.82)
  Dysphagia, Week 48: number analyzed (Participants) | 44 | 12
  Dysphagia, Week 48 | -5.30 (23.78) | 0.00 (14.21)
  Dysphagia, Week 57: number analyzed (Participants) | 36 | 8
  Dysphagia, Week 57 | -3.70 (29.58) | 4.17 (21.36)
  Dysphagia, Week 66: number analyzed (Participants) | 31 | 5
  Dysphagia, Week 66 | -6.45 (32.68) | 0.00 (0.00)
  Dysphagia, Week 75: number analyzed (Participants) | 25 | 4
  Dysphagia, Week 75 | -4.00 (27.76) | 16.67 (33.33)
  Dysphagia, Week 84: number analyzed (Participants) | 19 | 3
  Dysphagia, Week 84 | -8.77 (33.04) | 0.00 (0.00)
  Dysphagia, Week 93: number analyzed (Participants) | 20 | 2
  Dysphagia, Week 93 | 0.00 (28.61) | 0.00 (0.00)
  Dysphagia, Week 102: number analyzed (Participants) | 16 | 1
  Dysphagia, Week 102 | 0.00 (0.00) | 0.00 (NA) — The standard deviation is a measure of the amount of variation or dispersion of a set of values. Number analyzed is 1 so standard deviation is not available.
  Dysphagia, Week 111: number analyzed (Participants) | 14 | 0
  Dysphagia, Week 111 | -4.76 (22.10) |
  Dysphagia, Week 120: number analyzed (Participants) | 14 | 0
  Dysphagia, Week 120 | 2.38 (8.91) |
  Dysphagia, Week 129: number analyzed (Participants) | 14 | 0
  Dysphagia, Week 129 | -2.38 (20.52) |
  Dysphagia, Week 138: number analyzed (Participants) | 14 | 0
  Dysphagia, Week 138 | 4.76 (12.10) |
  Dysphagia, Week 147: number analyzed (Participants) | 14 | 0
  Dysphagia, Week 147 | -4.76 (28.81) |
  Dysphagia, Week 156: number analyzed (Participants) | 7 | 0
  Dysphagia, Week 156 | 0.00 (0.00) |
  Dysphagia, Week 165: number analyzed (Participants) | 8 | 0
  Dysphagia, Week 165 | -8.33 (23.57) |
  Dysphagia, Week 174: number analyzed (Participants) | 7 | 0
  Dysphagia, Week 174 | 0.00 (0.00) |
  Dysphagia, Week 183: number analyzed (Participants) | 4 | 0
  Dysphagia, Week 183 | 0.00 (0.00) |
  Dysphagia, Week 192: number analyzed (Participants) | 4 | 0
  Dysphagia, Week 192 | 0.00 (0.00) |
  Dysphagia, Week 201: number analyzed (Participants) | 2 | 0
  Dysphagia, Week 201 | 16.67 (23.57) |
  Dysphagia, Week 210: number analyzed (Participants) | 1 | 0
  Dysphagia, Week 210 | 0.00 (NA) — The standard deviation is a measure of the amount of variation or dispersion of a set of values. Number analyzed is 1 so standard deviation is not available. |
  Dysphagia, Safety Follow-Up Visit: number analyzed (Participants) | 11 | 13
  Dysphagia, Safety Follow-Up Visit | 12.12 (37.34) | 0.00 (19.25)
  Peripheral Neuropathy, Baseline: number analyzed (Participants) | 296 | 146
  Peripheral Neuropathy, Baseline | 11.26 (21.10) | 14.84 (24.46)
  Peripheral Neuropathy, Week 6: number analyzed (Participants) | 223 | 115
  Peripheral Neuropathy, Week 6 | 3.29 (19.74) | 1.45 (25.51)
  Peripheral Neuropathy, Week 12: number analyzed (Participants) | 151 | 64
  Peripheral Neuropathy, Week 12 | 1.99 (21.16) | 2.08 (26.48)
  Peripheral Neuropathy, Week 18: number analyzed (Participants) | 121 | 39
  Peripheral Neuropathy, Week 18 | 1.10 (19.21) | 5.13 (24.83)
  Peripheral Neuropathy, Week 24: number analyzed (Participants) | 106 | 30
  Peripheral Neuropathy, Week 24 | 3.77 (23.60) | 7.78 (22.63)
  Peripheral Neuropathy, Week 30: number analyzed (Participants) | 83 | 23
  Peripheral Neuropathy, Week 30 | 4.82 (20.25) | -1.45 (21.27)
  Peripheral Neuropathy, Week 36: number analyzed (Participants) | 60 | 16
  Peripheral Neuropathy, Week 36 | 7.78 (24.83) | 12.50 (29.50)
  Peripheral Neuropathy, Week 42: number analyzed (Participants) | 53 | 14
  Peripheral Neuropathy, Week 42 | 8.18 (23.48) | 9.52 (20.37)
  Peripheral Neuropathy, Week 48: number analyzed (Participants) | 44 | 12
  Peripheral Neuropathy, Week 48 | 6.82 (23.38) | 8.33 (20.72)
  Peripheral Neuropathy, Week 57: number analyzed (Participants) | 36 | 8
  Peripheral Neuropathy, Week 57 | 7.41 (25.34) | 20.83 (30.54)
  Peripheral Neuropathy, Week 66: number analyzed (Participants) | 32 | 5
  Peripheral Neuropathy, Week 66 | 6.25 (23.09) | 13.33 (38.01)
  Peripheral Neuropathy, Week 75: number analyzed (Participants) | 25 | 4
  Peripheral Neuropathy, Week 75 | 5.33 (22.93) | 8.33 (31.91)
  Peripheral Neuropathy, Week 84: number analyzed (Participants) | 19 | 3
  Peripheral Neuropathy, Week 84 | 8.77 (21.78) | 0.00 (0.00)
  Peripheral Neuropathy, Week 93: number analyzed (Participants) | 20 | 2
  Peripheral Neuropathy, Week 93 | 6.67 (17.44) | 0.00 (0.00)
  Peripheral Neuropathy, Week 102: number analyzed (Participants) | 16 | 1
  Peripheral Neuropathy, Week 102 | 6.25 (18.13) | 0.00 (NA) — The standard deviation is a measure of the amount of variation or dispersion of a set of values. Number analyzed is 1 so standard deviation is not available.
  Peripheral Neuropathy, Week 111: number analyzed (Participants) | 14 | 0
  Peripheral Neuropathy, Week 111 | 2.38 (15.82) |
  Peripheral Neuropathy, Week 120: number analyzed (Participants) | 14 | 0
  Peripheral Neuropathy, Week 120 | 2.38 (15.82) |
  Peripheral Neuropathy, Week 129: number analyzed (Participants) | 14 | 0
  Peripheral Neuropathy, Week 129 | 2.38 (15.82) |
  Peripheral Neuropathy, Week 138: number analyzed (Participants) | 14 | 0
  Peripheral Neuropathy, Week 138 | 0.00 (13.07) |
  Peripheral Neuropathy, Week 147: number analyzed (Participants) | 14 | 0
  Peripheral Neuropathy, Week 147 | 2.38 (15.82) |
  Peripheral Neuropathy, Week 156: number analyzed (Participants) | 7 | 0
  Peripheral Neuropathy, Week 156 | -4.76 (12.60) |
  Peripheral Neuropathy, Week 165: number analyzed (Participants) | 8 | 0
  Peripheral Neuropathy, Week 165 | 0.00 (17.82) |
  Peripheral Neuropathy, Week 174: number analyzed (Participants) | 7 | 0
  Peripheral Neuropathy, Week 174 | -4.76 (12.60) |
  Peripheral Neuropathy, Week 183: number analyzed (Participants) | 4 | 0
  Peripheral Neuropathy, Week 183 | -8.33 (16.67) |
  Peripheral Neuropathy, Week 192: number analyzed (Participants) | 4 | 0
  Peripheral Neuropathy, Week 192 | 16.67 (43.03) |
  Peripheral Neuropathy, Week 201: number analyzed (Participants) | 2 | 0
  Peripheral Neuropathy, Week 201 | 0.00 (0.00) |
  Peripheral Neuropathy, Week 210: number analyzed (Participants) | 1 | 0
  Peripheral Neuropathy, Week 210 | 0.00 (NA) — The standard deviation is a measure of the amount of variation or dispersion of a set of values. Number analyzed is 1 so standard deviation is not available. |
  Peripheral Neuropathy, Safety Follow-Up Visit: number analyzed (Participants) | 11 | 12
  Peripheral Neuropathy, Safety Follow-Up Visit | 21.21 (40.20) | -2.78 (33.21)
  Alopecia, Baseline: number analyzed (Participants) | 295 | 145
  Alopecia, Baseline | 7.91 (20.70) | 4.83 (15.70)
  Alopecia, Week 6: number analyzed (Participants) | 220 | 115
  Alopecia, Week 6 | -1.06 (19.48) | 6.09 (27.07)
  Alopecia, Week 12: number analyzed (Participants) | 149 | 63
  Alopecia, Week 12 | -2.01 (17.43) | 7.94 (27.90)
  Alopecia, Week 18: number analyzed (Participants) | 121 | 39
  Alopecia, Week 18 | -1.93 (17.90) | 12.82 (23.71)
  Alopecia, Week 24: number analyzed (Participants) | 105 | 28
  Alopecia, Week 24 | -1.27 (17.86) | 14.29 (30.67)
  Alopecia, Week 30: number analyzed (Participants) | 83 | 23
  Alopecia, Week 30 | -1.20 (19.79) | 10.14 (27.40)
  Alopecia, Week 36: number analyzed (Participants) | 60 | 16
  Alopecia, Week 36 | 5.56 (17.54) | 10.42 (29.11)
  Alopecia, Week 42: number analyzed (Participants) | 52 | 14
  Alopecia, Week 42 | 3.85 (14.24) | 7.14 (29.75)
  Alopecia, Week 48: number analyzed (Participants) | 43 | 12
  Alopecia, Week 48 | 3.10 (17.54) | 13.89 (36.12)
  Alopecia, Week 57: number analyzed (Participants) | 35 | 8
  Alopecia, Week 57 | 7.62 (18.23) | 29.17 (27.82)
  Alopecia, Week 66: number analyzed (Participants) | 30 | 5
  Alopecia, Week 66 | 6.67 (13.56) | 6.67 (14.91)
  Alopecia, Week 75: number analyzed (Participants) | 24 | 4
  Alopecia, Week 75 | 5.56 (12.69) | 8.33 (16.67)
  Alopecia, Week 84: number analyzed (Participants) | 19 | 3
  Alopecia, Week 84 | 1.75 (7.65) | 11.11 (19.25)
  Alopecia, Week 93: number analyzed (Participants) | 20 | 2
  Alopecia, Week 93 | 5.00 (12.21) | 16.67 (23.57)
  Alopecia, Week 102: number analyzed (Participants) | 16 | 1
  Alopecia, Week 102 | 4.17 (11.39) | 33.33 (NA) — The standard deviation is a measure of the amount of variation or dispersion of a set of values. Number analyzed is 1 so standard deviation is not available.
  Alopecia, Week 111: number analyzed (Participants) | 14 | 0
  Alopecia, Week 111 | 2.38 (8.91) |
  Alopecia, Week 120: number analyzed (Participants) | 14 | 0
  Alopecia, Week 120 | 4.76 (12.10) |
  Alopecia, Week 129: number analyzed (Participants) | 14 | 0
  Alopecia, Week 129 | 2.38 (8.91) |
  Alopecia, Week 138: number analyzed (Participants) | 14 | 0
  Alopecia, Week 138 | 7.14 (19.30) |
  Alopecia, Week 147: number analyzed (Participants) | 14 | 0
  Alopecia, Week 147 | 2.38 (8.91) |
  Alopecia, Week 156: number analyzed (Participants) | 7 | 0
  Alopecia, Week 156 | 0.00 (0.00) |
  Alopecia, Week 165: number analyzed (Participants) | 8 | 0
  Alopecia, Week 165 | 0.00 (0.00) |
  Alopecia, Week 174: number analyzed (Participants) | 7 | 0
  Alopecia, Week 174 | 0.00 (0.00) |
  Alopecia, Week 183: number analyzed (Participants) | 4 | 0
  Alopecia, Week 183 | 0.00 (0.00) |
  Alopecia, Week 192: number analyzed (Participants) | 4 | 0
  Alopecia, Week 192 | 8.33 (16.67) |
  Alopecia, Week 201: number analyzed (Participants) | 2 | 0
  Alopecia, Week 201 | 16.67 (23.57) |
  Alopecia, Week 210: number analyzed (Participants) | 1 | 0
  Alopecia, Week 210 | 0.00 (NA) — The standard deviation is a measure of the amount of variation or dispersion of a set of values. Number analyzed is 1 so standard deviation is not available. |
  Alopecia, Safety Follow-Up Visit: number analyzed (Participants) | 11 | 13
  Alopecia, Safety Follow-Up Visit | 0.00 (0.00) | 12.82 (44.18)
  Pain in Chest, Baseline: number analyzed (Participants) | 294 | 144
  Pain in Chest, Baseline | 20.29 (26.70) | 19.91 (24.72)
  Pain in Chest, Week 6: number analyzed (Participants) | 218 | 114
  Pain in Chest, Week 6 | -2.45 (26.66) | -4.09 (29.79)
  Pain in Chest, Week 12: number analyzed (Participants) | 149 | 63
  Pain in Chest, Week 12 | -4.03 (27.65) | -5.29 (31.80)
  Pain in Chest, Week 18: number analyzed (Participants) | 121 | 38
  Pain in Chest, Week 18 | -9.37 (27.29) | -5.26 (26.31)
  Pain in Chest, Week 24: number analyzed (Participants) | 105 | 29
  Pain in Chest, Week 24 | -7.62 (28.22) | -2.30 (28.07)
  Pain in Chest, Week 30: number analyzed (Participants) | 83 | 22
  Pain in Chest, Week 30 | -7.23 (31.26) | -9.09 (34.40)
  Pain in Chest, Week 36: number analyzed (Participants) | 60 | 14
  Pain in Chest, Week 36 | -11.67 (29.96) | 2.38 (30.56)
  Pain in Chest, Week 42: number analyzed (Participants) | 52 | 13
  Pain in Chest, Week 42 | -11.54 (34.86) | -2.56 (31.80)
  Pain in Chest, Week 48: number analyzed (Participants) | 43 | 11
  Pain in Chest, Week 48 | -17.83 (28.50) | 3.03 (17.98)
  Pain in Chest, Week 57: number analyzed (Participants) | 35 | 7
  Pain in Chest, Week 57 | -18.10 (30.62) | -4.76 (23.00)
  Pain in Chest, Week 66: number analyzed (Participants) | 31 | 4
  Pain in Chest, Week 66 | -15.05 (34.25) | -16.67 (19.25)
  Pain in Chest, Week 75: number analyzed (Participants) | 24 | 3
  Pain in Chest, Week 75 | -13.89 (21.80) | -22.22 (19.25)
  Pain in Chest, Week 84: number analyzed (Participants) | 19 | 2
  Pain in Chest, Week 84 | -22.81 (31.53) | -16.67 (23.57)
  Pain in Chest, Week 93: number analyzed (Participants) | 20 | 1
  Pain in Chest, Week 93 | -23.33 (26.71) | 0.00 (NA) — The standard deviation is a measure of the amount of variation or dispersion of a set of values. Number analyzed is 1 so standard deviation is not available.
  Pain in Chest, Week 102: number analyzed (Participants) | 16 | 0
  Pain in Chest, Week 102 | -20.83 (31.91) |
  Pain in Chest, Week 111: number analyzed (Participants) | 14 | 0
  Pain in Chest, Week 111 | -26.19 (29.75) |
  Pain in Chest, Week 120: number analyzed (Participants) | 14 | 0
  Pain in Chest, Week 120 | -26.19 (29.75) |
  Pain in Chest, Week 129: number analyzed (Participants) | 14 | 0
  Pain in Chest, Week 129 | -21.43 (21.11) |
  Pain in Chest, Week 138: number analyzed (Participants) | 14 | 0
  Pain in Chest, Week 138 | -26.19 (29.75) |
  Pain in Chest, Week 147: number analyzed (Participants) | 14 | 0
  Pain in Chest, Week 147 | -19.05 (36.31) |
  Pain in Chest, Week 156: number analyzed (Participants) | 7 | 0
  Pain in Chest, Week 156 | -23.81 (25.20) |
  Pain in Chest, Week 165: number analyzed (Participants) | 8 | 0
  Pain in Chest, Week 165 | -25.00 (23.57) |
  Pain in Chest, Week 174: number analyzed (Participants) | 7 | 0
  Pain in Chest, Week 174 | -23.81 (25.20) |
  Pain in Chest, Week 183: number analyzed (Participants) | 4 | 0
  Pain in Chest, Week 183 | -16.67 (33.33) |
  Pain in Chest, Week 192: number analyzed (Participants) | 4 | 0
  Pain in Chest, Week 192 | -16.67 (33.33) |
  Pain in Chest, Week 201: number analyzed (Participants) | 2 | 0
  Pain in Chest, Week 201 | -33.33 (47.14) |
  Pain in Chest, Week 210: number analyzed (Participants) | 1 | 0
  Pain in Chest, Week 210 | -66.67 (NA) — The standard deviation is a measure of the amount of variation or dispersion of a set of values. Number analyzed is 1 so standard deviation is not available. |
  Pain in Chest, Safety Follow-Up Visit: number analyzed (Participants) | 11 | 13
  Pain in Chest, Safety Follow-Up Visit | 0.00 (21.08) | 12.82 (21.68)
  Pain in Arm or Shoulder, Baseline: number analyzed (Participants) | 294 | 145
  Pain in Arm or Shoulder, Baseline | 19.16 (28.08) | 19.08 (27.43)
  Pain in Arm or Shoulder, Week 6: number analyzed (Participants) | 221 | 114
  Pain in Arm or Shoulder, Week 6 | -0.45 (26.87) | -0.58 (29.07)
  Pain in Arm or Shoulder, Week 12: number analyzed (Participants) | 149 | 63
  Pain in Arm or Shoulder, Week 12 | 0.67 (29.38) | -4.23 (30.81)
  Pain in Arm or Shoulder, Week 18: number analyzed (Participants) | 121 | 38
  Pain in Arm or Shoulder, Week 18 | -1.65 (30.08) | -2.63 (34.99)
  Pain in Arm or Shoulder, Week 24: number analyzed (Participants) | 104 | 28
  Pain in Arm or Shoulder, Week 24 | -3.21 (27.68) | 0.00 (28.69)
  Pain in Arm or Shoulder, Week 30: number analyzed (Participants) | 83 | 22
  Pain in Arm or Shoulder, Week 30 | -0.40 (26.80) | 4.55 (25.81)
  Pain in Arm or Shoulder, Week 36: number analyzed (Participants) | 60 | 15
  Pain in Arm or Shoulder, Week 36 | -4.44 (23.34) | -2.22 (34.43)
  Pain in Arm or Shoulder, Week 42: number analyzed (Participants) | 53 | 13
  Pain in Arm or Shoulder, Week 42 | -1.89 (25.67) | -5.13 (38.12)
  Pain in Arm or Shoulder, Week 48: number analyzed (Participants) | 44 | 11
  Pain in Arm or Shoulder, Week 48 | -1.52 (28.71) | -6.06 (35.96)
  Pain in Arm or Shoulder, Week 57: number analyzed (Participants) | 36 | 7
  Pain in Arm or Shoulder, Week 57 | 7.41 (25.34) | -9.52 (37.09)
  Pain in Arm or Shoulder, Week 66: number analyzed (Participants) | 31 | 4
  Pain in Arm or Shoulder, Week 66 | 1.08 (26.50) | -33.33 (38.49)
  Pain in Arm or Shoulder, Week 75: number analyzed (Participants) | 24 | 3
  Pain in Arm or Shoulder, Week 75 | -1.39 (26.88) | -33.33 (33.33)
  Pain in Arm or Shoulder, Week 84: number analyzed (Participants) | 19 | 2
  Pain in Arm or Shoulder, Week 84 | 3.51 (24.58) | -16.67 (23.57)
  Pain in Arm or Shoulder, Week 93: number analyzed (Participants) | 20 | 1
  Pain in Arm or Shoulder, Week 93 | 6.67 (23.20) | 0.00 (NA) — The standard deviation is a measure of the amount of variation or dispersion of a set of values. Number analyzed is 1 so standard deviation is not available.
  Pain in Arm or Shoulder, Week 102: number analyzed (Participants) | 16 | 0
  Pain in Arm or Shoulder, Week 102 | 8.33 (25.82) |
  Pain in Arm or Shoulder, Week 111: number analyzed (Participants) | 14 | 0
  Pain in Arm or Shoulder, Week 111 | 2.38 (27.62) |
  Pain in Arm or Shoulder, Week 120: number analyzed (Participants) | 14 | 0
  Pain in Arm or Shoulder, Week 120 | 4.76 (25.68) |
  Pain in Arm or Shoulder, Week 129: number analyzed (Participants) | 14 | 0
  Pain in Arm or Shoulder, Week 129 | 2.38 (27.62) |
  Pain in Arm or Shoulder, Week 138: number analyzed (Participants) | 14 | 0
  Pain in Arm or Shoulder, Week 138 | 2.38 (24.33) |
  Pain in Arm or Shoulder, Week 147: number analyzed (Participants) | 14 | 0
  Pain in Arm or Shoulder, Week 147 | 2.38 (27.62) |
  Pain in Arm or Shoulder, Week 156: number analyzed (Participants) | 7 | 0
  Pain in Arm or Shoulder, Week 156 | 9.52 (16.27) |
  Pain in Arm or Shoulder, Week 165: number analyzed (Participants) | 8 | 0
  Pain in Arm or Shoulder, Week 165 | 4.17 (11.79) |
  Pain in Arm or Shoulder, Week 174: number analyzed (Participants) | 7 | 0
  Pain in Arm or Shoulder, Week 174 | 0.00 (0.00) |
  Pain in Arm or Shoulder, Week 183: number analyzed (Participants) | 4 | 0
  Pain in Arm or Shoulder, Week 183 | 25.00 (31.91) |
  Pain in Arm or Shoulder, Week 192: number analyzed (Participants) | 4 | 0
  Pain in Arm or Shoulder, Week 192 | 0.00 (0.00) |
  Pain in Arm or Shoulder, Week 201: number analyzed (Participants) | 2 | 0
  Pain in Arm or Shoulder, Week 201 | 0.00 (0.00) |
  Pain in Arm or Shoulder, Week 210: number analyzed (Participants) | 1 | 0
  Pain in Arm or Shoulder, Week 210 | 0.00 (NA) — The standard deviation is a measure of the amount of variation or dispersion of a set of values. Number analyzed is 1 so standard deviation is not available. |
  Pain in Arm or Shoulder, Safety Follow-Up Visit: number analyzed (Participants) | 11 | 13
  Pain in Arm or Shoulder, Safety Follow-Up Visit | 12.12 (42.88) | 7.69 (33.76)
  Pain in other parts, Baseline: number analyzed (Participants) | 287 | 144
  Pain in other parts, Baseline | 25.32 (31.93) | 27.55 (31.86)
  Pain in other parts, Week 6: number analyzed (Participants) | 216 | 113
  Pain in other parts, Week 6 | -1.85 (29.05) | 1.18 (33.31)
  Pain in other parts, Week 12: number analyzed (Participants) | 147 | 62
  Pain in other parts, Week 12 | -0.91 (32.63) | -0.54 (34.93)
  Pain in other parts, Week 18: number analyzed (Participants) | 115 | 36
  Pain in other parts, Week 18 | -1.74 (36.63) | 11.11 (36.51)
  Pain in other parts, Week 24: number analyzed (Participants) | 104 | 28
  Pain in other parts, Week 24 | -3.53 (35.35) | -4.76 (38.18)
  Pain in other parts, Week 30: number analyzed (Participants) | 81 | 22
  Pain in other parts, Week 30 | -2.88 (38.08) | -7.58 (20.40)
  Pain in other parts, Week 36: number analyzed (Participants) | 59 | 15
  Pain in other parts, Week 36 | -5.08 (33.23) | 2.22 (29.46)
  Pain in other parts, Week 42: number analyzed (Participants) | 50 | 13
  Pain in other parts, Week 42 | -2.67 (33.56) | -12.82 (32.03)
  Pain in other parts, Week 48: number analyzed (Participants) | 43 | 11
  Pain in other parts, Week 48 | -4.65 (27.78) | -15.15 (34.52)
  Pain in other parts, Week 57: number analyzed (Participants) | 34 | 7
  Pain in other parts, Week 57 | -1.96 (34.76) | -9.52 (31.71)
  Pain in other parts, Week 66: number analyzed (Participants) | 29 | 4
  Pain in other parts, Week 66 | 3.45 (37.10) | -16.67 (43.03)
  Pain in other parts, Week 75: number analyzed (Participants) | 24 | 3
  Pain in other parts, Week 75 | 8.33 (31.47) | 0.00 (0.00)
  Pain in other parts, Week 84: number analyzed (Participants) | 19 | 2
  Pain in other parts, Week 84 | -1.75 (39.24) | 0.00 (0.00)
  Pain in other parts, Week 93: number analyzed (Participants) | 20 | 1
  Pain in other parts, Week 93 | -3.33 (28.41) | 0.00 (NA) — The standard deviation is a measure of the amount of variation or dispersion of a set of values. Number analyzed is 1 so standard deviation is not available.
  Pain in other parts, Week 102: number analyzed (Participants) | 16 | 0
  Pain in other parts, Week 102 | -4.17 (26.87) |
  Pain in other parts, Week 111: number analyzed (Participants) | 13 | 0
  Pain in other parts, Week 111 | -5.13 (29.96) |
  Pain in other parts, Week 120: number analyzed (Participants) | 14 | 0
  Pain in other parts, Week 120 | 0.00 (26.15) |
  Pain in other parts, Week 129: number analyzed (Participants) | 14 | 0
  Pain in other parts, Week 129 | -7.14 (14.19) |
  Pain in other parts, Week 138: number analyzed (Participants) | 14 | 0
  Pain in other parts, Week 138 | -7.14 (19.30) |
  Pain in other parts, Week 147: number analyzed (Participants) | 14 | 0
  Pain in other parts, Week 147 | 0.00 (18.49) |
  Pain in other parts, Week 156: number analyzed (Participants) | 7 | 0
  Pain in other parts, Week 156 | -14.29 (26.23) |
  Pain in other parts, Week 165: number analyzed (Participants) | 8 | 0
  Pain in other parts, Week 165 | -16.67 (25.20) |
  Pain in other parts, Week 174: number analyzed (Participants) | 7 | 0
  Pain in other parts, Week 174 | -9.52 (31.71) |
  Pain in other parts, Week 183: number analyzed (Participants) | 4 | 0
  Pain in other parts, Week 183 | 8.33 (63.10) |
  Pain in other parts, Week 192: number analyzed (Participants) | 4 | 0
  Pain in other parts, Week 192 | -8.33 (31.91) |
  Pain in other parts, Week 201: number analyzed (Participants) | 2 | 0
  Pain in other parts, Week 201 | -33.33 (0.00) |
  Pain in other parts, Week 210: number analyzed (Participants) | 1 | 0
  Pain in other parts, Week 210 | -66.67 (NA) — The standard deviation is a measure of the amount of variation or dispersion of a set of values. Number analyzed is 1 so standard deviation is not available. |
  Pain in other parts, Safety Follow-Up Visit: number analyzed (Participants) | 11 | 13
  Pain in other parts, Safety Follow-Up Visit | 9.09 (42.40) | 0.00 (33.33)

9. Secondary Outcome: Time to Deterioration (TTD) in Patient-Reported Lung Cancer Symptoms as Assessed by EORTC QLQ-C30 Score
Description: TTD with use of the EORTC was defined as the time from randomization to the first confirmed clinically meaningful deterioration in EORTC symptom scores. Confirmed clinically meaningful deterioration in lung cancer symptoms was defined as a = 10-point increase above baseline in a symptom score that must be held for at least two consecutive assessments or an initial = 10-point increase above baseline followed by either (a) death within 6 weeks from the last assessment through Week 48 or (b) death within 9 weeks from the last assessment from Week 48 thereafter. A = 10-point change in the EORTC scale score was perceived by participants as clinically significant (Osoba et al. 1998).
Time Frame: From baseline up to approximately 55 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Atezolizumab | Single Agent Chemotherapy (Vinorelbine or Gemcitabine)
Number analyzed (Participants) | 302 | 151
Months
  Dyspnoea | NA [19.0 to NA] — Median and/or CI are not estimable due to insufficient number of patients with events. | NA [8.3 to NA] — Median and/or CI are not estimable due to insufficient number of patients with events.
  Fatigue | 13.5 [8.3 to NA] — Median and/or CI are not estimable due to insufficient number of patients with events. | 8.4 [5.6 to NA] — Median and/or CI are not estimable due to insufficient number of patients with events.
Statistical Analysis 1: Comparison: Atezolizumab vs Single Agent Chemotherapy (Vinorelbine or Gemcitabine); Time to deterioration for Dyspnoea (single item QLQ-C30); Test type: Superiority — Stratified analysis. Histologic subtype, PD-L1 IHC status and brain metastases (Yes/No) were added as stratification factors; p = 0.975, Log Rank; Hazard Ratio (HR) = 1.01, 95% CI [0.57 to 1.78]
Statistical Analysis 2: Comparison: Atezolizumab vs Single Agent Chemotherapy (Vinorelbine or Gemcitabine); Time to deterioration for Fatigue (multi items QLQ-C30); Test type: Superiority — [test comment as in outcome 9, analysis 1]; p = 0.620, Log Rank; Hazard Ratio (HR) = 0.89, 95% CI 2-sided [0.55 to 1.42]

10. Secondary Outcome: TTD in Patient-Reported Lung Cancer Symptoms As Assessed by EORTC QLQ-LC13 Score
Description: TTD with use of the EORTC was defined as the time from randomization to the first confirmed clinically meaningful deterioration in EORTC symptom scores. Confirmed clinically meaningful deterioration in lung cancer symptoms was defined as a = 10-point increase above baseline in a symptom score that must be held for at least two consecutive assessments or an initial = 10-point increase above baseline followed by either (a) death within 6 weeks from the last assessment through Week 48 or (b) death within 9 weeks from the last assessment from Week 48 thereafter. A = 10-point change in the EORTC scale score was perceived by participants as clinically significant.
Time Frame: From baseline up to approximately 55 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Atezolizumab | Single Agent Chemotherapy (Vinorelbine or Gemcitabine)
Number analyzed (Participants) | 302 | 151
Months
  Cough | NA [NA to NA] — Median and/or CI are not estimable due to insufficient number of patients with events. | 21.4 [13.9 to NA] — Median and/or CI are not estimable due to insufficient number of patients with events.
  Chest Pain | NA [NA to NA] — Median and/or CI are not estimable due to insufficient number of patients with events. | NA [6.8 to NA] — Median and/or CI are not estimable due to insufficient number of patients with events.
  Dyspnoea | 17.3 [9.6 to 34.2] | 8.3 [5.5 to NA] — Median and/or CI are not estimable due to insufficient number of patients with events.
  Arm and/or Shoulder Pain | 21.3 [13.6 to NA] — Median and/or CI are not estimable due to insufficient number of patients with events. | 13.9 [8.6 to NA] — Median and/or CI are not estimable due to insufficient number of patients with events.
  Composite of Cough, Dyspnea and Chest Pain | 8.3 [5.5 to 17.3] | 4.2 [2.9 to 5.6]
Statistical Analysis 1: Comparison: Atezolizumab vs Single Agent Chemotherapy (Vinorelbine or Gemcitabine); Time to deterioration for Cough (single item QLQ-LC13); Test type: Superiority — [test comment as in outcome 9, analysis 1]; p = 0.653, Log Rank; Hazard Ratio (HR) = 1.16, 95% CI 2-sided [0.60 to 2.26]
Statistical Analysis 2: Comparison: Atezolizumab vs Single Agent Chemotherapy (Vinorelbine or Gemcitabine); Time to deterioration for Chest pain (single item QLQ-LC13); Test type: Superiority — [test comment as in outcome 9, analysis 1]; p = 0.036, Log Rank; Hazard Ratio (HR) = 0.51, 95% CI 2-sided [0.27 to 0.97]
Statistical Analysis 3: Comparison: Atezolizumab vs Single Agent Chemotherapy (Vinorelbine or Gemcitabine); Time to deterioration for Dyspnoea (multiple items QLQ-LC13); Test type: Superiority — [test comment as in outcome 9, analysis 1]; p = 0.125, Log Rank; Hazard Ratio (HR) = 0.70, 95% CI 2-sided [0.45 to 1.11]
Statistical Analysis 4: Comparison: Atezolizumab vs Single Agent Chemotherapy (Vinorelbine or Gemcitabine); Time to deterioration for Arm and/or shoulder pain (single item QLQ-LC13); Test type: Superiority — [test comment as in outcome 9, analysis 1]; p = 0.362, Log Rank; Hazard Ratio (HR) = 0.75, 95% CI 2-sided [0.41 to 1.39]
Statistical Analysis 5: Comparison: Atezolizumab vs Single Agent Chemotherapy (Vinorelbine or Gemcitabine); Time to Confirmed Deterioration for the Composite of the 3 following symptoms: cough, dyspnoea (multi-items QLQ-LC13) and chest pain; Test type: Superiority — [test comment as in outcome 9, analysis 1]; p = 0.041, Log Rank; Hazard Ratio (HR) = 0.68, 95% CI 2-sided [0.46 to 0.99]

11. Secondary Outcome: OS in Participants With Programmed Death-Ligand 1 (PD-L1) Positive Status
Description: OS was defined as the time between the date of randomization and the date of death due to any cause. OS was assessed in participants whose tumors express PD-L1 protein (i.e., tumor cell (TC) ≥1%) as measured by PD-L1 SP263 immunohistochemistry (IHC) assay. KM estimates were used to calculate the median.
Time Frame: From randomization up to death from any cause (up to approximately 55 months)
Population: ITT Population included all randomized participants irrespective of whether the assigned treatment was actually received. Overall number analyzed is the number of participants with data available for analysis.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Atezolizumab | Single Agent Chemotherapy (Vinorelbine or Gemcitabine)
Number analyzed (Participants) | 127 | 78
Months | 9.4 [7.0 to 11.3] | 10.3 [7.1 to 12.3]
Statistical Analysis 1: Comparison: Atezolizumab vs Single Agent Chemotherapy (Vinorelbine or Gemcitabine); SP263 TC>=1%; Test type: Superiority — [test comment as in outcome 9, analysis 1]; p = 0.272, Log Rank; Hazard Ratio (HR) = 0.84, 95% CI 2-sided [0.61 to 1.15]

12. Secondary Outcome: PFS as Determined by the Investigator Using RECIST v1.1 in Participants With PD-L1 Positive Status
Description: PFS was defined as the time from randomization to the first documented disease progression as determined by the investigator with the use of RECIST v1.1 or death from any cause, whichever occurs first. PD was defined as at least 20% increase in the sum of diameters of lesions, taking as reference the smallest sum during the study (nadir), including baseline. Investigator-assessed PFS was assessed in participants whose tumors express PD-L1 protein as measured by PD-L1 SP263 IHC assay. KM estimates were used to calculate the median.
Time Frame: as for outcome 3
Population: as for outcome 11
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Atezolizumab | Single Agent Chemotherapy (Vinorelbine or Gemcitabine)
Number analyzed (Participants) | 127 | 78
Months | 4.2 [2.9 to 5.8] | 3.0 [2.8 to 5.4]
Statistical Analysis 1: Comparison: Atezolizumab vs Single Agent Chemotherapy (Vinorelbine or Gemcitabine); SP263 TC>=1%; Test type: Superiority — [test comment as in outcome 9, analysis 1]; p = 0.366, Log Rank; Hazard Ratio (HR) = 0.87, 95% CI 2-sided [0.64 to 1.18]

ADVERSE EVENTS:
Time Frame: From Day 1 up to 90 days after last atezolizumab dose (up to approximately 62 months)
Description: Safety population included participants who received any amount of any study drug.
Arm/Group | Atezolizumab | Single Agent Chemotherapy (Vinorelbine or Gemcitabine)
All-Cause Mortality (participants affected / at risk) | 248/300 | 129/147
Serious Adverse Events (participants affected / at risk) | 147/300 | 54/147
Other Adverse Events (participants affected / at risk) | 234/300 | 128/147
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Atezolizumab (N=300) | Single Agent Chemotherapy (Vinorelbine or Gemcitabine) (N=147)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 3 (3)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Myelosuppression (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 2 (2)
Acute left ventricular failure (Cardiac disorders) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 2 (2) | 0 (0)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 3 (3) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac disorder (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 3 (3) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 1 (1) | 0 (0)
Myocarditis (Cardiac disorders) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (2) | 0 (0)
Diverticulum intestinal (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal toxicity (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small intestinal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Asthenia (General disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0)
Death (General disorders) | 7 (7) | 2 (2)
General physical health deterioration (General disorders) | 1 (1) | 1 (1)
Generalised oedema (General disorders) | 1 (1) | 0 (0)
Infusion site extravasation (General disorders) | 0 (0) | 1 (1)
Malaise (General disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0)
Oedema (General disorders) | 0 (0) | 1 (1)
Performance status decreased (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 3 (3) | 1 (1)
Sudden cardiac death (General disorders) | 2 (2) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Immune-mediated hepatitis (Hepatobiliary disorders) | 2 (2) | 0 (0)
Liver injury (Hepatobiliary disorders) | 1 (1) | 0 (0)
Systemic immune activation (Immune system disorders) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1)
Brain abscess (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 2 (2) | 1 (1)
COVID-19 (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 2 (2) | 0 (0)
Diarrhoea infectious (Infections and infestations) | 1 (1) | 0 (0)
Erysipelas (Infections and infestations) | 0 (0) | 1 (1)
Gastrointestinal infection (Infections and infestations) | 0 (0) | 1 (1)
Infectious pleural effusion (Infections and infestations) | 1 (1) | 0 (0)
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 5 (5) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 5 (5) | 4 (5)
Neutropenic sepsis (Infections and infestations) | 0 (0) | 2 (2)
Pneumonia (Infections and infestations) | 34 (38) | 11 (13)
Pneumonia aspiration (Infections and infestations) | 2 (2) | 0 (0)
Pneumonia bacterial (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia fungal (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia pneumococcal (Infections and infestations) | 1 (1) | 0 (0)
Relapsing fever (Infections and infestations) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 2 (2) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 4 (4)
Septic shock (Infections and infestations) | 2 (3) | 0 (0)
Skin infection (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 3 (3) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Femoral neck fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Radiation oesophagitis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Eastern Cooperative Oncology Group performance status worsened (Investigations) | 1 (1) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 2 (3) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 3 (7) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Fracture pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 2 (2)
Generalised tonic-clonic seizure (Nervous system disorders) | 1 (1) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 1 (1) | 0 (0)
Ischaemic cerebral infarction (Nervous system disorders) | 0 (0) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 0 (0)
Lacunar infarction (Nervous system disorders) | 1 (1) | 0 (0)
Lacunar stroke (Nervous system disorders) | 1 (1) | 0 (0)
Myasthenia gravis (Nervous system disorders) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 0 (0)
Spinal cord compression (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 2 (4) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 1 (1)
Confusional state (Psychiatric disorders) | 2 (2) | 0 (0)
Disorientation (Psychiatric disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 3 (3) | 2 (2)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 1 (1)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 2 (2)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Immune-mediated lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Laryngeal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 9 (10) | 2 (2)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 8 (9) | 2 (2)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (3)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Capillary leak syndrome (Vascular disorders) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 2 (2) | 0 (0)
Peripheral ischaemia (Vascular disorders) | 0 (0) | 1 (1)
Superior vena cava occlusion (Vascular disorders) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastroenteritis salmonella (Infections and infestations) | 1 (1) | 0 (0)
Klebsiella urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Periarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Iliac artery dissection (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Atezolizumab (N=300) | Single Agent Chemotherapy (Vinorelbine or Gemcitabine) (N=147)
Anaemia (Blood and lymphatic system disorders) | 50 (57) | 48 (70)
Leukopenia (Blood and lymphatic system disorders) | 3 (3) | 11 (15)
Neutropenia (Blood and lymphatic system disorders) | 2 (3) | 18 (39)
Hypothyroidism (Endocrine disorders) | 19 (22) | 0 (0)
Constipation (Gastrointestinal disorders) | 48 (61) | 28 (31)
Diarrhoea (Gastrointestinal disorders) | 40 (57) | 24 (45)
Nausea (Gastrointestinal disorders) | 32 (40) | 36 (54)
Vomiting (Gastrointestinal disorders) | 25 (33) | 23 (42)
Asthenia (General disorders) | 43 (49) | 19 (25)
Fatigue (General disorders) | 58 (74) | 34 (34)
Oedema peripheral (General disorders) | 25 (28) | 6 (6)
Pyrexia (General disorders) | 30 (35) | 10 (18)
Pneumonia (Infections and infestations) | 15 (15) | 5 (6)
Urinary tract infection (Infections and infestations) | 29 (47) | 12 (15)
Blood creatinine increased (Investigations) | 15 (26) | 4 (5)
Neutrophil count decreased (Investigations) | 2 (2) | 17 (26)
Weight decreased (Investigations) | 22 (30) | 11 (13)
White blood cell count decreased (Investigations) | 2 (2) | 15 (26)
Decreased appetite (Metabolism and nutrition disorders) | 66 (75) | 32 (40)
Hypokalaemia (Metabolism and nutrition disorders) | 18 (28) | 2 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 25 (28) | 7 (7)
Arthralgia (Musculoskeletal and connective tissue disorders) | 28 (36) | 12 (15)
Back pain (Musculoskeletal and connective tissue disorders) | 25 (29) | 13 (14)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 12 (12) | 8 (9)
Dizziness (Nervous system disorders) | 14 (18) | 8 (10)
Headache (Nervous system disorders) | 15 (20) | 7 (7)
Insomnia (Psychiatric disorders) | 17 (18) | 5 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 59 (72) | 13 (14)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 56 (60) | 14 (15)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 19 (26) | 9 (10)
Pruritus (Skin and subcutaneous tissue disorders) | 23 (34) | 3 (3)
Rash (Skin and subcutaneous tissue disorders) | 30 (44) | 5 (7)
Hypertension (Vascular disorders) | 23 (39) | 6 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2023-05-09): https://cdn.clinicaltrials.gov/large-docs/86/NCT03191786/Prot_002.pdf
  • Statistical Analysis Plan (2020-08-21): https://cdn.clinicaltrials.gov/large-docs/86/NCT03191786/SAP_001.pdf